

Title: A Randomized, Double-Blind, Double-Dummy, Parallel-group Phase 3 Study to Evaluate the Efficacy and Safety of Oral Once-Daily Administration of TAK-438 10 or 20 mg Compared to Lansoprazole 15 mg in the Maintenance Treatment of Subjects With Endoscopic Healing of Erosive Esophagitis

NCT Number: NCT02388737

SAP Approve Date: 08 January 2019

Certain information within this Statistical Analysis Plan has been redacted (ie, specific content is masked irreversibly from view with a black/blue bar) to protect either personally identifiable (PPD) information or company confidential information (CCI).

This may include, but is not limited to, redaction of the following:

- Named persons or organizations associated with the study.
- Proprietary information, such as scales or coding systems, which are considered confidential information under prior agreements with license holder.
- Other information as needed to protect confidentiality of Takeda or partners, personal information, or to otherwise protect the integrity of the clinical study.



1 of 58 **Template Number:** C-TMPL-DO-801 Page: **Version Number:** 1.0 **Effective Date:** 

This version replaces: **TMPL-104** 

**Template Title:** Statistical Analysis Plan (Legacy Takeda)

# TAKEDA DEVELOPMENT CENTER STATISTICAL ANALYSIS PLAN

STUDY NUMBER: TAK-438 305

the applicable reims of Use A Randomized, Double-Blind, Double-Dummy, Parallel-group Phase 3 Study to Evaluate the Efficacy and Safety of Oral Once-Daily Administration of TAK-438 10 or 20 mg Compared to Lansoprazole 15 mg in the Maintenance Treatment of Subjects With Endoscopic Healing of Erosive Esophagitis

Version: 2

Date: 08 January 2019

Property of Lakeda. For non-commercial Property of Lakeda.



C-TMPL-DO-801 **Template Number:**  **Version Number:** 1.0 **Effective Date:** 02 Apr 2014 Terms of Use

This version replaces: **TMPL-104** 

**Template Title:** Statistical Analysis Plan (Legacy Takeda)

#### 1.0 **APPROVAL SIGNATURES**

Electronic signatures can be found on the last page of this document.

A Randomized, Double-Blind, Double-Dummy, Parallel-group Phase 3 **Study Title:** 

Study to Evaluate the Efficacy and Safety of Oral Once-Daily C

Prodethy of Takeda. For noncommercial use only and subject to the Administration of TAK-438 10 or 20 mg Compared to Lansoprazole 15 mg in the Maintenance Treatment of Subjects With Endoscopic Healing of



Template Number: C-TMPL-DO-801  Version Number: 1.0 Effective Date: 02 Apr 2014

This version replaces: TMPL-104

Template Title: Statistical Analysis Plan (Legacy Takeda)

| 2.0 | TABLE OF CONTENTS | |
|---|---|---|
| 1.0 | APPROVAL SIGNATURES | 2 |
| 2.0 | TABLE OF CONTENTS | 3 |
| 3.0 | LIST OF ABBREVIATIONS | 6 |
| 4.0 | OBJECTIVES | 7 |
| 4.1 | PRIMARY OBJECTIVES | 7 |
| 4.2 | SECONDARY OBJECTIVES | 7 |
| 4.3 | ADDITIONAL OBJECTIVES | 7 |
| 4.4 | STUDY DESIGN | 7 |
| 5.0 | ANALYSIS ENDPOINTS | 9 |
| | Primary Endpoint | 9 |
| | Secondary Endpoint | 9 |
| | ADDITIONAL OBJECTIVES STUDY DESIGN ANALYSIS ENDPOINTS Primary Endpoint Secondary Endpoint Additional Endpoints DETERMINATION OF SAMPLE SIZE | 9 |
| 6.0 | DETERMINATION OF SAMPLE SIZE | . 10 |
| 7.0 | METHODS OF ANALYSIS AND PRESENTATION | . 11 |
| 7.1 | GENERAL CONSIDERATIONS. DEFINITIONS. | . 11 |
| 7.1.1 | DEFINITIONS | . 11 |
| 7.1.2 | DEFINITIONSANALYSIS SETS | |
| 7.1.3 | HANDLING OF RATE OF ENDOSCOPIC RECURRENCE OF EROSIVE ESOPHAGITIS | . 12 |
| 7.1.3.1 | Rate of Endoscopic Recurrence of Erosive Esophagitis During the first 12 Weeks of Treatment in the Maintenance Phase | 12 |
| 7.1.3.2 | Rate of Endoscopic Recurrence of Erosive Esophagitis During the 24-Week Maintenance Phase | . 12 |
| 7.1.4 | HANDLING OF DATA WHEN CALCULATING MEAN SEVERITY ACCORDING TO SUBJECT DIARY | 12 |
| 7.1.5 | HRQOL (EQ-5D-5L) | . 13 |
| 7.1.6 | HANDLING OF OTHER ENDPOINTS | |
| 7.2 | STUDY SUBJECTS, DEMOGRAPHICS, AND OTHER BASELINE CHARACTERISTICS | . 16 |
| 7.2.1.1<br>7.2.1.1 | DISPOSITION OF SUBJECTS | |
| 7.2.1.1 | Study Information | . 16 |
| 7.2.1.2 | Screen Failures | . 16 |
| 7.2.1.3 | Subject Eligibility | . 16 |
| 7.2.1.4 | Number of Subjects Randomized by Country, Site, and Treatment Group | . 17 |
| 7.2.1.5 | Disposition of Subjects | 17 |



C-TMPL-DO-801 4 of 58 **Template Number:** Page: **Version Number:** 1.0 **Effective Date:** 02 Apr 2014

| Version Number: 1.0 Effective Date: 02 Apr 2014 This version replaces: TMPL-104 Template Title: Statistical Analysis Plan (Legacy Takeda) | | |
|---|---|---|
| | Protocol Deviations and Analysis Sets | |
| 7.2.1.0 | | 18~5 |
| | Protocol Deviations Analysis Sets | 4.6218 |
| 7.2.2 | DEMOGRAPHICS AND OTHER BASELINE CHARACTERISTICS | 18 |
| 7.2.2.1 | DEMOGRAPHICS AND OTHER BASELINE CHARACTERISTICS Summary of Demographics and Other Baseline Characteristics Medical History and Concurrent Medical Conditions Medication History and Concomitant Medications TREATMENT COMPLIANCE | 18 |
| 7.2.2.2 | Medical History and Concurrent Medical Conditions | 19 |
| 7.2.2.3 | Medication History and Concomitant Medications. | 20 |
| 7.2.3 | TREATMENT COMPLIANCE | 20 |
| 7.2.3.1 | Study Drug Exposure and Compliance | 20 |
| 7.3 | EFFICACY ANALYSIS | 21 |
| 7.3.1 | PRIMARY EFFICACY ENDPOINT | 21 |
| 7.3.1.1 | Primary Analysis. | 21 |
| 7.3.1.2 | Secondary Analysis | 21 |
| 7.3.2 | EFFICACY ANALYSIS PRIMARY EFFICACY ENDPOINT Primary Analysis Secondary Analysis SECONDARY EFFICACY ENDPOINT | 21 |
| 7.3.2.1 | Rate of Endoscopic Recurrence of Erosive Esophaguis During the First 12 Weeks of Treatment in the Maintenance Phase | ie<br>21 |
| 7.3.2.2 | Sensitivity Analysis. | 22 |
| 7.3.3 | ADDITIONAL EFFICACY ENDPOINTS | 22 |
| 7.3.3.1 | Gastrointestinal Symptoms Based on Subject Diary | 22 |
| | Heartburn Symptoms | 22 |
| | Gastric Acid Regurgitation | 22 |
| 7.3.3.2 | HRQoL (EQ-5D-5L) | |
| | EQ-5D-5L Index Value | 23 |
| | EQ VAS Score | 24 |
| 7.3.3.3 | Barrett's Mucosa | |
| 7.3.4 | STATISTICAL/ANALYTICAL ISSUES | 24 |
| 7.3.4.1 | Adjustments for Covariates | 24 |
| 7.3.4.2 | Handling of Dropouts or Missing Data | 24 |
| 7.3.4.3 | Interim Analyses and Data Monitoring | |
| 7.3.4.4 | Multicenter Studies | |
| 7.3.4.5 | Multiple Comparison/Multiplicity | |
| 7.3.4.6 | Use of an "Efficacy Subset" of Subjects | |
| 7.3.4.7 | Active-Control Studies Intended to Show Equivalence or Non-Inferiority | |
| 7.3.4.8 | Subgroup Analysis | 26 |




This version replaces: TMPL-104

Template Title: Statistical Analysis Plan (Legacy Takeda)

| 7.4 | SAFETY ANALYSIS | |
|---|---|---|
| 7.4.1 | TREATMENT-EMERGENT ADVERSE EVENTS | 27 |
| 7.4.1.1 | Overview of Treatment-Emergent Adverse Events. | .02 |
| 7.4.1.2 | Displays of Treatment-Emergent Adverse Events | 28 |
| 7.4.2 | PRETREATMENT EVENTS AND ADVERSE EVENTS IN THE HEALING PHASE | 30 |
| 7.4.2.1 | Displays of Treatment-Emergent Adverse Events PRETREATMENT EVENTS AND ADVERSE EVENTS IN THE HEALING PHASE Displays of Pretreatment Events Displays of Adverse Events in the Healing Phase LABORATORY AND OTHER SAFETY DATA | 30 |
| 7.4.2.2 | Displays of Adverse Events in the Healing Phase. | 30 |
| 7.4.3 | LABORATORY AND OTHER SAFETY DATA | 31 |
| 7.4.3.1 | Laboratory Test Results. | 3 |
| | Hematology and Serum Chemistry | 31 |
| | LABORATORY AND OTHER SAFETY DATA Laboratory Test Results. Hematology and Serum Chemistry Urinalysis. Serum Gastrin, Pepsinogen I/II. | 32 |
| | Serum Gastrin, Pepsinogen I/II | 32 |
| 7.4.4 | - VITAL SICING PRINCIPLAL PUNDUNCIS AND OTREK UNSSEK VALIONS KELATED TO SAFET | 1 7 |
| | Vital Signs | 33 |
| | Vital Signs 12-lead ECG SUBGROUP ANALYSIS FOR CHINA SUBGROUP ANALYSIS FOR TAIWAN | 33 |
| 7.4.5 | SUBGROUP ANALYSIS FOR CHINA | 34 |
| 7.4.6 | SUBGROUP ANALYSIS FOR TAIWANS | 34 |
| 7.4.7 | SUBGROUP ANALYSIS FOR SAFETY ANALYSIS SET EXCLUDING ACCIDENTALLY UNBLINDED SUBJECTS | 34 |
| 7.4.8 | SIGNIFICANCE LEVEL AND CONFIDENCE COEFFICIENT | 34 |
| 7.4.9 | CHANGES IN THE STATISTICAL ANALYSIS PLAN | 35 |
| 8.0 | REFERENCES | 54 |
| 9.0 | APPENDIX | 55 |
| 9.1 | CRITERIA FOR MARKEDLY ABNORMAL VALUES | 5: |
| 9.1.1 | HEMATOLOGY, SERUM CHEMISTRY, URINALYSIS, VITAL SIGNS, AND 12-LEAD ECG (EXCEPT UPPER MAV CRITERIA OF QTCF INTERVAL) | 5: |
| 9.1.2 | 12-LEAD ECG (UPPER MAV CRITERIA OF QTCF INTERVAL) | |
| 9.2 | CRITERIA FOR ELEVATED LIVER ENZYME | |



6 of 58 **Template Number:** C-TMPL-DO-801 Page: to the applicable reims of Use applicable reims of Use **Version Number:** 1.0 **Effective Date:** 

This version replaces: **TMPL-104** 

**Template Title:** Statistical Analysis Plan (Legacy Takeda)

#### 3.0 LIST OF ABBREVIATIONS

AΕ adverse event

ALT alanine aminotransferase ALP alkaline phosphatase **ANCOVA** analysis of covariance **AST** aspartate aminotransferase

**BMI** body mass index **BUN** blood urea nitrogen Cochran-Mantel-Haenszel **CMH CPK** creatine phosphokinase **ECG** electrocardiogram

the 5-level version of the EuroQOL five dimensions questionnaire EQ-5D-5L

full analysis set **FAS GGT** γ-glutamyl transferase H. pylori Helicobacter pylori

Health-Related Quality of Life **HRQoL** LA classification Los Angeles classification LDH lactate dehydrogenase LLN lower limit of normal least square means LS means

MAV markedly abnormal value

Medical Dictionary for Regulatory Activities MedDRA mixed model repeated measures analysis **MMRM** 

proton pump inhibitor PPI PPS per protocol set QOL quality-of-life

Fridericia's corrected QT QTcF SAP statistical analysis plan

Tbili total bilirubin

**TEAE** treatment-emergent adverse event

ULN upper limit of normal

WHO Drug World Health Organization Drug Dictionary

WMWodds Wilcoxon-Mann-Whitney odds



C-TMPL-DO-801 7 of 58 **Template Number:** Page: 1.0 **Version Number: Effective Date:** 02 Apr 2014 reins of Use

This version replaces: **TMPL-104** 

**Template Title:** Statistical Analysis Plan (Legacy Takeda)

#### 4.0 **OBJECTIVES**

#### 4.1 PRIMARY OBJECTIVES

To demonstrate the non-inferiority of TAK-438 to Lansoprazole in the reduction of relapse of erosive esophagitis in subjects in the Maintenance Phase (24 weeks) in whom endoscopic healing of erosive esophagitis has been confirmed after treatment with TAK-438 or a PPI.

To determine the clinically recommended dose of TAK-438 for maintenance therapy in erosive esophagitis in whom endoscopic healing of erosive esophagitis has been confirmed after treatment with TAK-438 or a PPI.

#### 4.2 **SECONDARY OBJECTIVES**

- To evaluate the efficacy of TAK-438 during the first 12-weeks of treatment in the Maintenance Phase in subjects with endoscopically confirmed healed erosive esophagitis receiving TAK-438 or a PPI.
- To evaluate the safety of TAK-438 versus Lansoprazole in subjects in the Maintenance Phase (24 weeks) in whom endoscopic healing of erosive esophagitis has been confirmed after treatment with TAK-438 or a PPI.

#### **ADDITIONAL OBJECTIVES** 4.3

To evaluate the effect of TAK-438 on subjective symptoms of erosive esophagitis (heartburn and regurgitation) and improvement in Health Related Quality of Life using the EuroQol (EQ-5D-5L).

#### 4.4 STUDY DESIGN

This is a phase 3, multicenter, randomized double-blind, parallel-group study to demonstrate the non-inferiority of TAK-438 (10 mg or 20 mg) to Lansoprazole 15 mg in preventing the recurrence of erosive esophagitis in subjects with endoscopically confirmed healing of erosive esophagitis. This study also aims to determine the clinically recommended dose of TAK-438 for maintenance therapy of erosive esophagitis.

This study is comprised of 2 treatment periods: An open-label, single-arm period in which subjects receive Lansoprazole 30 mg for up to 8 weeks (Healing Phase), and a double-blind, parallel-group period in which subjects are randomized at a 1:1:1 ratio to TAK-438 10 mg, 20 mg or Lansoprazole 15 mg once daily for up to 24 weeks (Maintenance Phase). To entoil in the study subjects must have ongoing erosive esophagitis or have completed Study TAK-438 303. Subjects with ongoing erosive esophagitis are required to undergo the Healing Phase. Once erosive esophagitis healing is confirmed by endoscopy, these subjects may be randomized to 1 of 3 treatments in the Maintenance Phase. Subjects with endoscopic-confirmed healing of erosive esophagitis following the completion of Study TAK-438 303 will be randomized into the Maintenance Phase without carrying out the open-label Healing Phase. Subjects who previously entered the study (prior to Protocol Amendment 06) after confirmation of healed erosive esophagitis following treatment with a proton pump inhibitor (termed "de novo" subjects) are no longer eligible to enter the study; any ongoing subjects may continue being treated in the Maintenance Phase. A schematic of the study design is included in Figure 4.a.

If relapse of erosive esophagitis has been endoscopically confirmed in any subject, the subject will complete the study at that time point (to be construed as "complete cases in the Maintenance Phase"), regardless of the time point where relapse of disease is confirmed.

This study will be conducted at a total of around 70 sites across Asia with an estimated total of 231 subjects randomized to each treatment group during the Maintenance Phase (totaling 693 subjects entering the Maintenance Phase for the study).



Template Number: C-TMPL-DO-801 
Version Number: 1.0 Effective Date: 02 Apr 2014

This version replaces: TMPL-104

Template Title: Statistical Analysis Plan (Legacy Takeda)

The study will consist of a Screening Phase of up to 28 days duration (Visit 1), a Healing Phase (for those subjects with ongoing erosive esophagitis only) of 4 or 8 weeks duration (Visits 2<sub>HP</sub> and 3<sub>HP</sub>), followed by a Maintenance Phase of up to 24 weeks (Visits 2-8), and a Follow-up Period of up to 14 days duration. With the exception of the Follow-up (which will be carried out by phone), all visits will occur at the clinic. The total duration of treatment is up to 6 months (24 weeks) in subjects entering from Study TAK-438\_303, and up to 8 months (32 weeks) in subjects entering the study with ongoing erosive esophagitis.

Subjects with ongoing erosive esophagitis: Subjects who have ongoing erosive esophagitis will enter the Healing Phase and administration of Lansoprazole 30 mg once daily will commence following the completion of all required assessments at Visit 2<sub>HP</sub>. Subjects will then undergo a visit at Week -4 (Visit 3<sub>HP</sub>), where the subject may undergo endoscopy to confirm healing of erosive esophagitis. This is an optional procedure where the decision to perform endoscopy is based on the investigator's clinical judgment of a subject's symptoms of healing. Subjects who do not show endoscopic healing at Visit 3<sub>HP</sub> may continue in the Healing Phase and undergo endoscopy at Day 1 (Visit 2). Subjects with endoscopically confirmed healing of erosive esophagitis at Week -4 or at Day 1 will be eligible to enter the Maintenance Phase. Where the results from clinical laboratory tests confirming eligibility for the Maintenance Phase at Week -4 are not immediately available, subjects should continue to receive Lansoprazole 30 mg for up to 14 days. Subjects healed at Day 1 should be immediately randomized. Subjects who do not have endoscopic-confirmed healed erosive esophagitis after 8 weeks treatment (Healing Phase Failures) will not be randomized into the Maintenance Phase and should be treated using routine clinical care.

Subjects with healed erosive esophagitis: Subjects with healed erosive esophagitis will undergo a randomization visit (Visit 2), and dosing for the Maintenance Phase will commence following the completion of all required assessments on Day 1. Visits will then occur at 2 week intervals after the initiation of treatment in the Maintenance Phase. As a result of Protocol Amendment 06, subjects with healed erosive esophagitis following treatment with a proton pump inhibitor outside Study TAK-438\_303 or the Healing Phase of the current study (*de novo* subjects) are no longer eligible to enter the study; any ongoing subjects may continue to be treated in the Maintenance Phase.

All subjects receiving TAK-438 must undergo a total of 8 weeks of LFT monitoring visits with visits occurring every 2 weeks. For subjects entering the Maintenance Phase of the current study within 7 days of completing Study TAK-438 303, the requirement for 8 weeks of monitoring can be totalled across the 2 studies.



Figure 4.a Schematic of Study Design



**Template Number:** C-TMPL-DO-801 9 of 58 Page: **Version Number:** 1.0 reims of Use **Effective Date:** 02 Apr 2014

This version replaces: **TMPL-104** 

**Template Title:** Statistical Analysis Plan (Legacy Takeda)

#### 5.0 **ANALYSIS ENDPOINTS**

#### Primary Endpoint

The primary efficacy endpoint for this study is the rate of recurrence\* of erosive esophagitis as confirmed on endoscopy during the 24-week Maintenance Phase.

\*Recurrence: defined as subjects endoscopically confirmed to have erosive esophagitis (LA classification grades A to D) during the Maintenance Phase (24 weeks).

### Secondary Endpoint

The secondary efficacy endpoint for this study is the rate of recurrence\* of erosive esophagitis during the first 12 weeks of treatment in the Maintenance Phase. Safety endpoints for this study include adverse events (AEs), clinical laboratory test results, ECG, vital signs, serum gastrin and pepsinogen I/II levels

\*Recurrence: defined as subjects endoscopically confirmed to have erosive esophagitis (LA classification grades A to D) during the Maintenance Phase (12 weeks).

#### Additional Endpoints

Other efficacy endpoints include subjective symptoms of erosive esophagitis (heartburn and regurgitation) as recorded in subject diaries and Health-Related Quality of Life measures.

Property of Takeda. For non-commercial use of enality of Link



10 of 58 **Template Number:** C-TMPL-DO-801 Page: **Version Number:** 1.0 02 Apr 2014 **Effective Date:** 

Assuming that the true Week 24 recurrence rate is 30.4% for Lansoprazole, 22.0% for TAK-438 10 mg, and 13.6% for TAK-438 20 mg, and assuming that the dropout rate is approximately 30%, a sample size of 208 subjects per group will provide an overall power of 90% to establish non-inferiority using a 2-sided 95% or non-inferiority margin. 231 subjects per group will be included to 11 requirements of various countries

The assumption of the true recurrence rate is based on a phase 3 study that showed a Week 24 recurrence rate of 30.4% for Lansoprazole 15 mg and 13.6% for Lansoprazole 30 mg.

Frogaty of Takeda. For non-commercial use only and subject to Based on results from an earlier study of Lansoprazole as maintenance therapy for erosive esophagitis (AG-1749/CCT-202), the point estimate for the difference (Lansoprazole 15 mg group—famotidine group) was calculated as -57.6% with the upper limit of the confidence interval being -30.7%. Therefore, the non-inferiority



C-TMPL-DO-801 11 of 58 **Template Number:** Page: **Version Number:** 1.0 **Effective Date:** 02 Apr 2014 ible Leiths of Use

This version replaces: **TMPL-104** 

**Template Title:** Statistical Analysis Plan (Legacy Takeda)

#### METHODS OF ANALYSIS AND PRESENTATION 7.0

#### 7.1 GENERAL CONSIDERATIONS

#### 7.1.1 **Definitions**

The following definitions and calculation formulas will be used.

- TEAE: An adverse event whose date of onset occurs on or after the start of the Maintenance Phase drug. A TEAE whose relationship to the Maintenance Phase drug is missing will be considered drug-related. A TEAE whose intensity is missing will be considered severe.
- Descriptive statistics: number of subjects, mean, standard deviation, maximum, minimum, and quartiles
- Study Day: The day before the first dose of the Maintenance Phase drug will be defined as Study Day -1 and the day of the first dose will be defined as Study Day 1. Other study days are defined relative to Study Day 1, eg, the day prior to Study Day 1 is Day -1 and the day after Study Day 1 is Day 2.
- Follow-up Day: The day after the last dose of the Maintenance Phase drug will be defined as Follow-up Day 1. Other follow-up days are defined relative to Follow-up Day 1.
- Duration of exposure to study drug (days): date of last dose of Maintenance Phase drug date of first dose of Maintenance Phase drug + 1.
- Study drug compliance (%): (number of days the subject answered "Yes" in the subject diary to the question "Study medication taken?") / duration of exposure to study drug \* 100 (rounded to 1 decimal place).
- Age (years): The following only applies to subjects from countries other than Korea. If the date informed consent obtained or the date of birth is missing, then age will be missing. If the month and the day of the date informed consent obtained is before the month and the day of the date of birth, then age will be calculated as follows: the year of the date informed consent obtained - the year of the date of birth - 1. For all others, age will be calculated as follows: the year of the date informed consent obtained - the year of the date of birth.
- BMI (kg/m<sup>2</sup>): weight (kg) / (height (m))<sup>2</sup> (rounded to 1 decimal place).
- Pepsinogen I/II Ratio: Pepsinogen I (μg/L) / Pepsinogen II (μg/L) (rounded to 1 decimal place).
  - QTcF interval (msec). QT interval (msec) / (RR interval (sec)) $^{0.33}$  (rounded to the nearest whole number).
  - Confidence interval for one sample proportion: Exact (Clopper-Pearson) confidence interval will be used.
  - Confidence interval for two sample proportion difference: Wald confidence interval will be used.
- Significant TEAE: Any TEAE (not including serious TEAEs) that led to an intervention, including withdrawal of drug treatment, dose increase, dose reduction, or significant additional concomitant therapy.

### **Analysis Sets**

Analysis of efficacy variables will be conducted in the full analysis set (FAS) defined as all randomized subjects who receive at least 1 dose of the Maintenance Phase drug and have at least 1 post-baseline endoscopy, and will be based on the randomized treatment. Randomized subjects who were accidentally unblinded due to IWRS system error will be excluded.

The primary efficacy endpoint and the secondary efficacy endpoint will also be analyzed in the per protocol set defined as all FAS subjects who did not have any of the major protocol deviations listed below. Analyses will be based on the randomized treatment.



C-TMPL-DO-801 12 of 58 **Template Number:** Page: **Version Number:** 1.0 **Effective Date:** 02 Apr 2014 ible Letins of Use

This version replaces: **TMPL-104** 

**Template Title:** Statistical Analysis Plan (Legacy Takeda)

- Subjects who did not meet inclusion criteria #3 or #4
- Subjects who met exclusion criteria #8, #11, #12, #13, or #14
- Subjects with study drug compliance of less than 70%
- Subjects who have been unblinded prior to database lock
- Subjects who have violated the rules specified in section 7.3 of the protocol

Analysis of safety variables will be conducted in the safety analysis set defined as all subjects who take at least 1 dose of the Maintenance Phase drug and will be based on the treatment received in the Maintenance Phase.

#### Handling of Rate of Endoscopic Recurrence of Erosive Esophagitis 7.1.3

## 7.1.3.1 Rate of Endoscopic Recurrence of Erosive Esophagitis During the first 12 Weeks of Treatment in the Maintenance Phase

A subject who is diagnosed as LA classification grade A, B, C, or D from endoscopy tests performed between Study Day 2 and Study Day 127 (up to and including Follow-up Day 14) will be considered as a relapsed subject. Subjects who do not have any endoscopy data during this period will be treated as missing. Subjects who do not meet this requirement will be considered as 'not relapsed'. Recurrence rate will be calculated from the relapsed and not relapsed subjects, however, any subjects diagnosed as LA classification grade A, B, C, or D from endoscopy tests performed before the Maintenance Phase drug administration will be excluded from the analysis.

# 7.1.3.2 Rate of Endoscopic Recurrence of Erosive Esophagitis During the 24-Week Maintenance Phase

A subject who is diagnosed as LA classification grade A, B, C, or D from endoscopy tests performed after Study Day 2 (up to and including Follow-up Day 14) will be considered as a relapsed subject. Subjects who do not have any endoscopy data during this period will be treated as missing. Subjects who do not meet this requirement will be considered as 'not relapsed'. Recurrence rate will be calculated from the relapsed and not relapsed subjects, however, any subjects diagnosed as LA classification grade A, B, C, or D from endoscopy tests performed before the Maintenance Phase drug administration will be excluded from the analysis.

#### Handling of Data When Calculating Mean Severity According to Subject 7.1.4 Diary

Each subjective symptom of erosive esophagitis as recorded in subject diaries (ie, heartburn, gastric acid regurgitation) will be handled as below.

Severity will be scored as follows. None: 0, Mild: 1, Moderate: 2, Severe: 3.

For each subject, the mean severity will be calculated as follows at each visit. If the denominator is missing, then the calculated result should also be missing.

Mean severity = (total score of the severity recorded for the visit) / (number of days the severity of symptom is recorded) (rounded to 2 decimal places)

(Note: Severity recorded as "Not Completed" will be treated as missing.)

The following visits will be used.



**Template Number:** C-TMPL-DO-801  able reims of Use **Version Number:** 1.0 **Effective Date:** 

This version replaces: **TMPL-104** 

**Template Title:** Statistical Analysis Plan (Legacy Takeda)

| Visit | Time Interval (days) | |
|-----------|----------------------|-------------------------------------|
| VISIL | Study Day | Follow-up Day |
| Baseline* | Day -6 – Day 1 | |
| Week 4 | Day 2 – Day 29 | up to and including Follow-up Day 1 |
| Week 8 | Day 30 – Day 57 | up to and including Follow-up Day 1 |
| Week 12 | Day 58 – Day 85 | up to and including Follow-up Day |
| Week 16 | Day 86 – Day 113 | up to and including Follow-up Day I |
| Week 20 | Day 114 – Day 141 | up to and including Follow-up Day 1 |
| Week 24 | Day 142 – Day 169 | up to and including Follow-up Day 1 |

<sup>\*:</sup> Will not be included in the analysis, however, data will be created.

#### 7.1.5 HRQoL (EQ-5D-5L)

All evaluable data (ie, non-missing) obtained in the corresponding time interval will be used in evaluating the EQ-5D-5L index value and EQ VAS score. If more than one observation lies within the same visit window, the observation with the closest Study Day to the scheduled Study Day will be used. If there are two observations equidistant to the scheduled Study Day, the later observation will be used.

The EQ-5D-5L index values will be calculated from the EQ-5D-5L descriptive system scores based on the EQ-5D-5L Crosswalk value sets. If any of the questions are not answered, the EQ-5D-5L index value of the day will be treated as missing.

The following visits will be used.

| | Visit Schedule | | | Time Interval (days) |
|---|---|---|---|---|
| | VISIt | (days) | Study Day | Follow-up Day |
| | Baseline | Study Day: 1 | -28 – 1 | |
| | Week 4 | Study Day: 29 | 2 – 57 | up to and including Follow-up Day 14 |
| | Week 12 | Study Day: 85 | 58 – 127 | up to and including Follow-up Day 14 |
| | Week 24 | Study Day: 169 | 128 – 211 | up to and including Follow-up Day 14 |
| Property | Katega. | | | |




For each visit, all evaluable observation (ie, non-missing) obtained in the corresponding time interval will be used. If more than one observation lies within the same visit window, the observation with the closest Study Day to the scheduled Study Day will be used. If there are two observations equidistant to the scheduled Study Day will be used.

The following visits will be used.

Weight, BMI, Endoscopy (esophageal hiatal hernia)

| Visit | Scheduled Study Day (days) | Time Interval (days) | |
|---|---|---|---|
| | | Study Day | Follow-up Day |
| Baseline | Study Day: 1 | up to and including Study Day 1 | |
| Endoscopy (Barrett's mucosa), 12-lead ECG | | | |

| | Endoscopy (Barrett's mucosa), 12-lead ECG | | | |
|---|---|---|---|---|
| | Visit Scheduled Study Day Time Interval (days) Study Day Fol | | | nterval (days) |
| | VISIt | (days) | Study Day | Follow-up Day |
| | Baseline | Study Day: | up to and including Study Day 1 | |
| | Week 12 | Study Day: 85 | 2 – 127 | up to and including<br>Follow-up Day 14 |
| | Week 24 | Study Day: 169 | 128 – 211 | up to and including<br>Follow-up Day 14 |
| Property | Week 24 | | | |



Template Number: C-TMPL-DO-801 

This version replaces: TMPL-104

Template Title: Statistical Analysis Plan (Legacy Takeda)

Clinical laboratory tests (ALT, AST, total bilirubin, and direct bilirubin)

| Visit | Scheduled Study Day | Time Interval (days) | |
|---|---|---|---|
| VISIL | (days) | Study Day | Follow-up Day |
| Baseline* | Study Day: 1 | -28 – 1 | . (2) |
| Week 2 | Study Day: 15 | 2 – 22 | up to and including<br>Follow-up Day 14 |
| Week 4 | Study Day 29 | 23 – 36 | up to and including<br>Follow-up Day 14 |
| Week 6 | Study Day: 43 | 37 – 50 | up to and including<br>Follow-up Day 14 |
| Week 8 | Study Day: 57 | 51-71 | up to and including<br>Follow-up Day 14 |
| Week 12 | Study Day: 85 | 72 – 127 | up to and including<br>Follow-up Day 14 |
| Week 24 | Study Day: 169 | 128 – 211 | up to and including<br>Follow-up Day 14 |

<sup>\*:</sup> For the clinical laboratory tests of the subjects who participated in the TAK-438\_303 study, if the last study visit coincides with the first visit in the 305 study or if the subject was randomized in the 305 study within 7 days after completing the last visit in the 303 study, then the data obtained at the last visit can be used as the baseline data for the 305 study.

Clinical laboratory tests (other than ALT, AST, total bilirubin, and direct bilirubin), Gastrin, Pepsinogen I/II, Vital signs

| Visit | Scheduled Study Day | Time Interval (days) | |
|---|---|---|---|
| VISIT | (days) | Study Day | Follow-up Day |
| Baseline* | Study Day: 1 | -28 – 1 | |
| Week 4 | Study Day 29 | 2 – 57 | up to and including<br>Follow-up Day 14 |
| Week 12 | Study Day: 85 | 58 – 127 | up to and including<br>Follow-up Day 14 |
| Week 24 | Study Day: 169 | 128 – 211 | up to and including<br>Follow-up Day 14 |

\*: For the clinical laboratory tests, gastrin, and pepsinogen I/II of the subjects who participated in the TAK-438\_303 study, if the last study visit coincides with the first visit in the 305 study or if the subject was randomized in the 305 study within 7 days after completing the last visit in the 303 study, then the data obtained at the last visit can be used as the baseline data for the 305 study.



**Template Number:** C-TMPL-DO-801 16 of 58 Page: to the applicable Terms of Use on w **Version Number:** 1.0 **Effective Date:** 02 Apr 2014

This version replaces: **TMPL-104** 

**Template Title:** Statistical Analysis Plan (Legacy Takeda)

#### 7.2 STUDY SUBJECTS, DEMOGRAPHICS, AND OTHER BASELINE CHARACTERISTICS

#### 7.2.1 **Disposition of Subjects**

#### 7.2.1.1 Study Information

Analysis Set: All Subjects Who Signed the Informed Consent Form Analysis Variables: Date First Subject Signed Informed Consent Form

Date of Last Subject's Last Visit/Contact

MedDRA Version WHO Drug Version

SAS Version Used for Creating the Datasets

Analytical Methods: (1) Study Information

Study information shown in the analysis variables section will be provided.

#### 7.2.1.2 Screen Failures

All Subjects Who Were Not Randomized? Analysis Set:

 $[Min \le -.. < 65, 65 \le -.. < 75, 75 \le -.. \le Max]$ Analysis Variables: Age (years)

> Gender [Male, Female]

Race [American Indian or Alaska Native, Asian, Black or African American,

Native Hawaiian or Other Pacific Islander, White, Multiple]

Analytical Methods: (1) Screen Failures

Frequency distributions for categorical variables and descriptive statistics for continuous

variables will be provided.

# 7.2.1.3 Subject Eligibility

All Subjects Who Signed the Informed Consent Form Analysis Set:

Eligibility Status Analysis Variables: [Yes, No]

Primary Reason for Subject Not Being Eligible [Pretreatment Event/Adverse Event,

> Major Protocol Deviation, Lost to Follow-Up, Voluntary Withdrawal,

Study Termination,

Did Not Meet Entrance Criteria,

Healing Phase Failure,

Other]

Analytical Methods: (1) Eligibility for Randomization

> Frequency distributions will be provided. When calculating the percentages for the primary reasons for subject not being eligible, the total number of ineligible subjects will

be used as the denominator.



**Template Number:** C-TMPL-DO-801 17 of 58 Page: **Version Number:** 1.0 **Effective Date:** 02 Apr 2014 he Letins of Use

This version replaces: **TMPL-104** 

**Template Title:** Statistical Analysis Plan (Legacy Takeda)

### 7.2.1.4 Number of Subjects Randomized by Country, Site, and Treatment Group

Randomized Set Analysis Set:

Analysis Variables: Randomization Status [Yes]

Stratum: [China, Malaysia, South Korea, Taiwan] Country

> Site [Site numbers will be used as categories]

(1) Number of Subjects Randomized by Country, Site, and Treatment Group Analytical Methods:

Frequency distribution will be provided for each stratum by treatment group and overall. to the 312

### 7.2.1.5 Disposition of Subjects

Randomized Set Analysis Set:

Analysis Variables: Maintenance Phase Drug Administration [No]

Status

Reason for Not Being Treated [Pretreatment Event/Adverse Event,

Major Protocol Deviation, Lost to Follow-Up,

Voluntary Withdrawal, Study Termination,

Pregnancy, Lack of Efficacy, Other]

Maintenance Phase Drug Completion Status [Completed Maintenance Phase Drug,

Prematurely Discontinued Maintenance Phase

Reason for Discontinuation of Maintenance [Pretreatment Event/Adverse Event,

Phase Drug Major Protocol Deviation, Lost to Follow-Up,

> Voluntary Withdrawal, Study Termination, Pregnancy, Lack of Efficacy, Other]

(1) Disposition of Subjects Analytical Methods:

> Frequency distributions will be provided for each treatment group and overall. When calculating percentages for the reasons for not being treated, the total number of subjects not treated by the maintenance phase drug will be used as the denominator. When calculating percentages for the reasons for discontinuation of maintenance phase drug, the total number of subjects who prematurely discontinued the maintenance phase drug will be used as the denominator.

Property of Takedai. For (2) Flow Chart of Subject Distribution

Flow chart will be provided.



**Template Number:** C-TMPL-DO-801  **Version Number:** 1.0 **Effective Date:** 02 Apr 2014 Who Leithe of Use

This version replaces: **TMPL-104** 

**Template Title:** Statistical Analysis Plan (Legacy Takeda)

#### 7.2.1.6 Protocol Deviations and Analysis Sets

#### **Protocol Deviations**

Analysis Set: Randomized Set

[Entry Criteria, Concomitant Medication, Analysis Variables: Protocol Deviation

Procedure Not Performed Per Protocol

Study Medication, Withdrawal Criterial

Analytical Methods: (1) Protocol Deviations

> Frequency distribution will be provided by treatment group and overall for each deviation category. A subject who has several deviations will be counted once in each appropriate category. A subject who has several deviations that can be classified into the same ind subject

category will be counted only once.

**Analysis Sets** 

Analysis Set: Randomized Set Analysis Variables: Analysis Sets

Full Analysis Set [Included] Per Protocol Set [Included] [Included] Safety Analysis Set

Analytical Methods:

(1) Analysis Sets

Frequency distributions will be provided by treatment group and overall.

#### **Demographics and Other Baseline Characteristics** 7.2.2

# 7.2.2.1 Summary of Demographics and Other Baseline Characteristics

Analysis Set: Randomized Set

Full Analysis Set

Analysis Variables: Country [China, Malaysia, South Korea, Taiwan] Property of Lakedai.

Participation in TAK-438 303 Study [Yes, No]

Age (years)  $[Min \le -.. \le 65, 65 \le -.. \le 75, 75 \le -.. \le Max]$ 

Gender [Male, Female]

Race [American Indian or Alaska Native, Asian,

Black or African American.

Native Hawaiian or Other Pacific Islander,

White, Multiple]

Min<= - <150, 150<= - <160, Height (cm)

 $160 \le -170, 170 \le -180$ 

Weight (kg) (Baseline)  $[Min \le - <50.0, 50.0 \le - <60.0,$ 

 $60.0 \le -80.0$ ,  $70.0 \le -80.0$ ,

 $80.0 \le - \le Max$ 



**Template Number:** C-TMPL-DO-801 19 of 58 Page: **Version Number:** 1.0 **Effective Date:** 02 Apr 2014 Terms of Use

This version replaces: **TMPL-104** 

**Template Title:** Statistical Analysis Plan (Legacy Takeda)

> BMI (kg/m<sup>2</sup>) (Baseline) Min<= - <18.5, 18.5<= - <25.0,

> > $25.0 \le - \le Max$

[The Subject Has Never Smoked, Smoking Classification

The Subject Is a Current Smoker,

The Subject Is an Ex-smoker]

Consumption of Alcohol [Drink Everyday,

> Drink a Couple of Days Per Week Drink a Couple of Days Per Month,

Never Drink]

Consumption of Caffeine [Yes, No]

[Yes (End of Treatment: Within the Past 1 Year), History of H. pylori Eradication Yes (End of Treatment: More than 1 Year), No] Therapy

[Grade A, Grade B, Grade C, Grade D] LA Classification (Time of Diagnosis)

[Grade A/B, Grade C/D]

[Present (3 cm or Greater), Barrett's Mucosa (Baseline)

Present (Less than 3 cm), Absent, Unknown]

Present (2 cm or Greater), Esophageal Hiatal Hernia (Baseline)

Present (Less than 2 cm), Absent, Unknown]

HRQoL (EQ-5D-5L)

EQ-5D-5L Index Value (Baseline)

EQ VAS Score (Baseline)

Analytical Methods:

(1) Summary of Demographics and Other Baseline Characteristics

Frequency distributions for categorical variables and descriptive statistics for continuous

variables will be provided by treatment group and overall.

### 7.2.2.2 Medical History and Concurrent Medical Conditions

Analysis Set:

Safety Analysis Set

Analysis Variables:

Medical History

Concurrent Medical Conditions

Analytical Methods:

(1) Medical History by System Organ Class and Preferred Term

(2) Concurrent Medical Conditions by System Organ Class and Preferred Term

Frequency distributions will be provided for each treatment group. MedDRA dictionary

will be used for coding. Summaries will be provided using SOC and PT, where SOC

will be sorted alphabetically and PT will be sorted in decreasing frequency.

A subject with multiple occurrences of medical history or concurrent medical condition

within a SOC will be counted only once in that SOC. A subject with multiple

occurrences of medical history or concurrent medical condition within a PT will be

counted only once in that PT.




**TMPL-104** This version replaces:

**Template Title:** Statistical Analysis Plan (Legacy Takeda)

### 7.2.2.3 Medication History and Concomitant Medications

Analysis Set: Safety Analysis Set Analysis Variables: Medication History

**Concomitant Medications** 

Analytical Methods: (1) Medication History by Preferred Medication Name

licable terms of Use (2) Concomitant Medications That Started Prior to and Were Ongoing at Baseline as well as Those That Started After Baseline by Preferred Medication Name Frequency distributions will be provided for each treatment group. WHO Drug dictionary will be used for coding. Summaries will be provided using preferred medication names and sorted in decreasing frequency based on the number of reports. A subject who has been administered several medications with the same preferred medication name will be counted only once for that preferred medication name.

#### 7.2.3 **Treatment Compliance**

# 7.2.3.1 Study Drug Exposure and Compliance

Analysis Set: Safety Analysis Set

 $[Min \le - <50.0, 50.0 \le - <70.0,$ 

 $70.0 \le - 90.0, 90.0 \le - = Max$ 

Frequency distributions for categorical variables and descriptive statistics for



**Template Number:** C-TMPL-DO-801 21 of 58 Page: **Version Number:** 1.0 **Effective Date:** 02 Apr 2014

This version replaces: **TMPL-104** 

**Template Title:** Statistical Analysis Plan (Legacy Takeda)

#### 7.3 **EFFICACY ANALYSIS**

insofuse The full analysis set will be the main analysis set used. The per protocol set will be used for analyses performed secondarily on the primary efficacy endpoint and secondary efficacy endpoints in order to examine the robustness of the results.

#### 7.3.1 **Primary Efficacy Endpoint**

#### 7.3.1.1 Primary Analysis

Analysis Set: Full Analysis Set

Rate of Endoscopic Recurrence of Erosive Esophagitis During the 24-week Maintenance Analysis Variable:

Phase (%)

(1) Rate of Endoscopic Recurrence of Erosive Esophagitis During the 24-week Analytical Methods:

**Maintenance Phase** 

Frequency distributions will be provided by treatment group along with rates and the two-sided 95% confidence intervals. The differences in the rates between each TAK-438 group and the Lansoprazole group (each TAK-438 group – the Lansoprazole group) and the two-sided 95% confidence intervals using the Wald method will be provided. The non-inferiority margin will be set to 10%. Details concerning interpretation are described

in section 7.3.4.5.

#### 7.3.1.2 Secondary Analysis

Analysis Set: Per Protocol Set

Rate of Endoscopic Recurrence of Erosive Esophagitis During the 24-week Maintenance Analysis Variable:

Phase (%)

(1) Sensitivity Analysis Analytical Methods:

To check the robustness of the results, the same analyses as those in section 7.3.1.1 will

be performed using the per protocol set.

#### Secondary Efficacy Endpoint 7.3.2

## 7.3.2.1 Rate of Endoscopic Recurrence of Erosive Esophagitis During the First 12 Weeks of Treatment in the Maintenance Phase

Analysis Set: Full Analysis Set

Analysis Variable: Rate of Endoscopic Recurrence of Erosive Esophagitis During the First 12 Weeks of

Treatment in the Maintenance Phase (%)

Analytical Methods: (1) Rate of Endoscopic Recurrence of Erosive Esophagitis During the First 12 Weeks of

Treatment in the Maintenance Phase

Frequency distributions will be provided by treatment group along with rates and the two-sided 95% confidence intervals. The differences in the rates between each TAK-438 group and the Lansoprazole group (each TAK-438 group – the Lansoprazole group) and

the two-sided 95% confidence intervals will also be provided.



C-TMPL-DO-801 22 of 58 Template Number: Page: **Version Number:** 1.0 **Effective Date:** 02 Apr 2014 (eims of Use

This version replaces: **TMPL-104** 

**Template Title:** Statistical Analysis Plan (Legacy Takeda)

#### 7.3.2.2 Sensitivity Analysis

Analysis Set: Per Protocol Set

Rate of Endoscopic Recurrence of Erosive Esophagitis During the First 12 Weeks of Analysis Variable:

Treatment in the Maintenance Phase (%)

Analytical Methods: (1) Sensitivity Analysis

To check the robustness of the results, the same analyses as section 7.3.2.1 will be

performed using the per protocol set.

#### 7.3.3 **Additional Efficacy Endpoints**

# 7.3.3.1 Gastrointestinal Symptoms Based on Subject Diary

#### Heartburn Symptoms

Analysis Set: Full Analysis Set

Mean Severity of Symptoms Analysis Variables: Subgroups: Barrett's Mucosa (Baseline)

Visit: Week 4, Week 8, Week 12, Week 16, Week 20, Week 24

The following summaries will be provided for each treatment group. Analytical Methods:

Descriptive statistics will be provided for each visit.

The difference in the medians between each TAK-438 group and the Lansoprazole ii) group (each TAK-438 group – the Lansoprazole group) and the two-sided 95% confidence intervals will be provided for each visit using the Hodges-Lehmann

estimator. Wilcoxon rank-sum tests will be used to test for treatment differences at each

visit.

iii) WMWodds of each TAK-438 group to the Lansoprazole group and the two-sided 95% confidence intervals will be provided for each visit based on Wilcoxon-Mann-Whitney test statistics.

#### Subgroup Analysis (Baseline Barrett's Mucosa)

The same analyses as all of the above will be conducted for the defined subgroups.

#### Gastric Acid Regurgitation

Analysis Set: Full Analysis Set

Analytical Methods: The same analyses as those in section 7.3.3.1 "Heartburn Symptoms" will be conducted for

the gastric acid regurgitation.



C-TMPL-DO-801 23 of 58 **Template Number:** Page: **Version Number:** 1.0 **Effective Date:** 02 Apr 2014

This version replaces: **TMPL-104** 

**Template Title:** Statistical Analysis Plan (Legacy Takeda)

### 7.3.3.2 HRQoL (EQ-5D-5L)

#### EQ-5D-5L Index Value

Analysis Set: Full Analysis Set Analysis Variables: EQ-5D-5L Index Value

Covariates: LA Classification (Time of Diagnosis)

> EQ-5D-5L Index Value (Baseline) Baseline, Week 4, Week 12, Week 24

Visit: Analytical Methods: (1) Summary of EQ-5D-5L Index Value

[Grade A/B, Grade C/D]; and the for the Descriptive statistics will be provided for each visit for the observed values and for each post-baseline visit for the changes from baseline (each post-baseline visit - baseline) by treatment group. The mean differences in the changes from baseline between each TAK-438 group and the Lansoprazole group (each TAK-438 group – the Lansoprazole group) and the two-sided 95% confidence intervals will be provided for each post-baseline visit. Two sample t-tests will be used to test for treatment differences at each post-baseline visit.

#### (2) ANCOVA

The changes from baseline (each post baseline visit - baseline) in the analysis variable will be analyzed using an ANCOVA model with treatment and LA classification at the time of diagnosis as factors and baseline EQ-5D-5L index value as a covariate. The ANCOVA analysis will be performed at each post baseline visit. LS means and the twosided 95% confidence intervals will be provided for each treatment group. The difference in the LS means between each TAK-438 group and the Lansoprazole group (each TAK-438 group – the Cansoprazole group) and the two-sided 95% confidence interval will be provided. The difference in the LS means will be tested for treatment differences.

#### (3) MMRM

Property of Lakeda: Fork

The changes from baseline (each post baseline visit – baseline) in the analysis variable will be analyzed using a mixed model repeated measures analysis (MMRM) model with the changes from baseline in the analysis variable as the response, and treatment, LA classification at the time of diagnosis, baseline value of the analysis variable, visit, treatment-by-visit interaction, baseline-by-visit interaction, and LA grade-by-visit interaction as fixed effects. LS means and the two-sided 95% confidence intervals will be provided by visit for each treatment group. The differences in the LS means between each TAK-438 group and the Lansoprazole group (each TAK-438 group - the Lansoprazole group) and the two-sided 95% confidence intervals will be provided for each visit. The differences in the LS means will be tested for treatment differences. An unstructured variance-covariance matrix will be used to model the within-subject errors and Satterthwaite's method will be used to approximate the degrees of freedom.



**Template Number:** C-TMPL-DO-801 24 of 58 Page: **Effective Date: Version Number:** 1.0 02 Apr 2014 ible Leiths of Use

This version replaces: **TMPL-104** 

**Template Title:** Statistical Analysis Plan (Legacy Takeda)

#### **EQ VAS Score**

Analysis Set: Full Analysis Set Analysis Variables: EQ VAS Score

Covariates: LA Classification (Time of Diagnosis) [Grade A/B, Grade C/D]

EQ VAS Score (Baseline)

The same analyses as those in section 7.3.3.2 "EQ-5D-5L Index Value" will be conducted for Analytical Methods:

the EQ VAS score.

#### 7.3.3.3 Barrett's Mucosa

Analysis Set: Full Analysis Set

[Increased, Unchanged, Reduced, Disappeared, Unknown] Analysis Variables: Barrett's Mucosa (Change) [Present (3 cm or Greater), Present (Less than 3 cm), Absent, Subgroups: Barrett's Mucosa (Baseline)

Unknown]

Visit: Week 12, Week 24

Analytical Methods: (1) Frequency distribution of Barrett's Mucosa (Change) by Baseline Barrett's Mucosa

Frequency distribution will be provided for each subgroup and visit by treatment group.

#### Statistical/Analytical Issues 7.3.4

# 7.3.4.1 Adjustments for Covariates

Analysis Set: Full Analysis Set

Rate of Endoscopic Recurrence of Erosive Esophagitis During the 24-week Maintenance Analysis Variable:

Phase (%)

Rate of Endoscopic Recurrence of Erosive Esophagitis During the First 12 Weeks of

Treatment in the Maintenance Phase (%)

Stratified Variable: LA Classification (Time of Diagnosis) [Grade A/B, Grade C/D]

(1) CMH Test for the Rate of Endoscopic Recurrence of Erosive Esophagitis During the Analytical Methods:

24-week Maintenance Phase

(2) CMH Test for the Rate of Endoscopic Recurrence of Erosive Esophagitis During the First 12 Weeks of Treatment in the Maintenance Phase

A CMH test with LA Classification at the time of diagnosis as a stratification factor will be used to compare the above analysis variable between each TAK-438 group and the Lansoprazole group for treatment differences. Mantel-Haenszel estimate of risk difference between each TAK-438 group and the Lansoprazole group (each TAK-438 group – the Lansoprazole group) and the two-sided 95% confidence interval using the

Wald method will also be provided.

#### 7.3.4.2 Handling of Dropouts or Missing Data

For the primary endpoint "rate of endoscopic recurrence of erosive esophagitis during the 24-week maintenance phase" and the secondary efficacy endpoint "rate of endoscopic recurrence of erosive esophagitis during the first 12



C-TMPL-DO-801 **Template Number:** 25 of 58 Page: **Version Number:** 1.0 **Effective Date:** 02 Apr 2014

Values below the lower limit of quantification will be treated as zero when calculating the descriptive statistics.

Values above the upper limit of quantification will be treated as the upper limit values when calculating the descriptive statistics.

7.3.4.3 Interim Analyses and 5 ect to the applicable

No interim analysis is planned in this study.

#### 7.3.4.4 Multicenter Studies

Treatment-by-center interaction will not be explored in this study.

### 7.3.4.5 Multiple Comparison/Multiplicity

Adjustment for multiplicity will be performed for the primary endpoint "rate of endoscopic recurrence of erosive esophagitis during the 24-week maintenance phase" and the secondary efficacy endpoint "rate of endoscopic recurrence of erosive esophagitis during the first 12 weeks of treatment in the maintenance phase" in the following order under the closed testing procedure and the analysis will be conducted using the full analysis set.

- The primary endpoint "rate of endoscopic recurrence of erosive esophagitis during the 24-week maintenance phase" will be tested for non-inferiority between the TAK-438 20 mg group and the Lansoprazole group. In other words, if the upper bound of the 95% confidence interval of the treatment difference (the TAK-438 20 mg group) the Lansoprazole group) is ≤10%, the non-inferiority for TAK-438 20 mg relative to Lansoprazole will be declared.
- If the previous test is successful, the primary endpoint will be tested for non-inferiority between the TAK-438 10 mg group and the Lansoprazole group. In other words, if the upper bound of the 95% confidence interval of the treatment difference (the TAK-438 10 mg group – the Lansoprazole group) is ≤10%, the non-inferiority for TAK-438 10 mg relative to Lansoprazole will be declared.
- If the previous test is successful, the primary endpoint will be tested for superiority between the TAK-438 20 mg group and the Lansoprazole group. The upper bound of the 95% confidence interval of the treatment difference (the TAK-438 20 mg group -the Lansoprazole group) will be compared to 0%.
- If the previous test is successful, the primary endpoint will be tested for superiority between the TAK-438 10 mg group and the Lansoprazole group.
- If the previous test is successful, the secondary endpoint "rate of endoscopic recurrence of erosive esophagitis during the first 12 weeks of treatment in the maintenance phase" will be tested for superiority between the TAK-438 20 mg group and the Lansoprazole group.
- If the previous test is successful, the secondary endpoint will be tested for superiority between the TAK-438 10 mg group and the Lansoprazole group.



**Template Number:** C-TMPL-DO-801 26 of 58 Page: **Version Number:** 1.0 **Effective Date:** 02 Apr 2014

This version replaces: **TMPL-104** 

**Template Title:** Statistical Analysis Plan (Legacy Takeda)

reins of Use Other analyses in this study will be done only for exploratory purposes and multiplicity adjustments will not be made.

### 7.3.4.6 Use of an "Efficacy Subset" of Subjects

In addition to analyses on the primary and secondary efficacy endpoints using the full analysis set, sensitivity analyses will also be performed using the per protocol set to examine the robustness of the results.

# 7.3.4.7 Active-Control Studies Intended to Show Equivalence or Non-Inferiority

For the primary efficacy endpoint, non-inferiority for each TAK-438 group relative to the Lansoprazole group will be confirmed in the full analysis set using a non-inferiority margin of 10%.

# 7.3.4.8 Subgroup Analysis

Analysis Set: Full Analysis Set

Rate of Endoscopic Recurrence of Erosive Esophagitis During the 24-week Maintenance Analysis Variable:

Phase (%)

Rate of Endoscopic Recurrence of Erosive Esophagitis During the First 12 Weeks of

Treatment in the Maintenance Phase (%)

 $[Min \le -.. \le 65, 65 \le -.. \le 75, 75 \le -.. \le Max]$ Subgroups: Age (years)

Gender [Male, Female]

BMI (kg/m<sup>2</sup>) (Baseline)  $[Min \le -.. < 18.5, 18.5 \le -.. < 25.0, 25.0 \le -.. \le Max]$ 

LA Classification (Time of Diagnosis) [Grade A/B, Grade C/D]

Barrett's Mucosa (Baseline) [Present, Absent]

Esophageal Hiatal Hernia (Baseline) [Present (2 cm or Greater),

Present (Less than 2 cm), Absent, Unknown]

Analytical Methods: (1) Subgroup Analysis for the Rate of Endoscopic Recurrence of Erosive Esophagitis Property of Takedai. For no **During the 24-week Maintenance Phase** 

(2) Subgroup Analysis for the Rate of Endoscopic Recurrence of Erosive Esophagitis During the First 12 Weeks of Treatment in the Maintenance Phase

The same analyses as those in section 7.3.1.1 will be performed for each of the above subgroups, except for non-inferiority testing.



**Template Number:** C-TMPL-DO-801 27 of 58 Page: applicable Terms of Use **Version Number:** 1.0 **Effective Date:** 02 Apr 2014

This version replaces: **TMPL-104** 

**Template Title:** Statistical Analysis Plan (Legacy Takeda)

#### 7.4 SAFETY ANALYSIS

#### 7.4.1 Treatment-Emergent Adverse Events

#### 7.4.1.1 Overview of Treatment-Emergent Adverse Events

Analysis Set: Safety Analysis Set

Analysis Variables: **TEAE** 

Categories: Relationship to Study Drug [Related, Not Related]

> [Mild, Moderate, Severe] Intensity

Analytical Methods: The following summaries will be provided for each treatment group

#### (1) Overview of Treatment-Emergent Adverse Events

- 1) All Treatment-Emergent Adverse Events (number of events, number and percentage of subjects)
- 2) Relationship of Treatment-Emergent Adverse Events to Study Drug (number of events, number and percentage of subjects)
- 3) Intensity of Treatment-Emergent Adverse Events (number of events, number and percentage of subjects)
- 4) Treatment-Emergent Adverse Events Leading to Study Drug Discontinuation (number of events, number and percentage of subjects)
- 5) Relationship to Study Drug of Treatment-Emergent Adverse Events Leading to Study Drug Discontinuation (number of events, number and percentage of subjects)
- 6) Serious Treatment-Emergent Adverse Events (number of events, number and percentage of subjects)
- 7) Relationship of Serious Treatment-Emergent Adverse Events to Study Drug (number of events, number and percentage of subjects)
- 8) Serious Treatment-Emergent Adverse Events Leading to Study Drug Discontinuation (number of events, number and percentage of subjects)
- (9) Treatment-Emergent Adverse Events Resulting in Death (number of events, number and percentage of subjects)
- 10) Treatment-Emergent Adverse Events Corresponding to Liver Function Test Abnormalities (number of events, number and percentage of subjects)
- 11) Significant Treatment-Emergent Adverse Events (number of events, number and percentage of subjects)

Property of Takedai. For TEAEs will be counted according to the rules below.

#### Number of subjects

Summaries for 2), 5), and 7)

A subject with occurrences of TEAE in both categories (ie, Related and Not Related) will be counted once in the Related category.

Summary for 3)

A subject with multiple occurrences of TEAE will be counted once for the TEAE with the maximum intensity.



C-TMPL-DO-801 28 of 58 Template Number: Page: in the series of 1.0 **Version Number: Effective Date:** 02 Apr 2014

This version replaces: **TMPL-104** 

**Template Title:** Statistical Analysis Plan (Legacy Takeda)

Summaries other than 2), 3), 5), and 7)

A subject with multiple occurrences of TEAE will be counted only once.

Number of events

For each summary, the total number of events will be calculated.

#### 7.4.1.2 Displays of Treatment-Emergent Adverse Events

Analysis Set: Safety Analysis Set

Analysis Variables: **TEAE** 

Property of Takedai.

[Mild, Moderate, Severe] Categories: Intensity

> $[1 \le - \le 84, 85 \le - \le 168, 169 \le - \le Max]$ Time of Onset (day)

Analytical Methods: The following summaries will be provided using frequency distribution for each treatment

group.

TEAEs will be coded using the MedDRA and will be summarized using SOC and PT. SOC will be sorted alphabetically and PT will be sorted in decreasing frequency for tables provided by SOC and PT. SOC and PT will be sorted in decreasing frequency for tables provided by SOC only or PT only.

- (1) Treatment-Emergent Adverse Events by System Organ Class and Preferred Term
- (2) Treatment-Emergent Adverse Events by System Organ Class
- (3) Treatment-Emergent Adverse Events by Preferred Term
- (4) Drug-Related Treatment-Emergent Adverse Events by System Organ Class and Preferred Term
- (5) Intensity of Treatment-Emergent Adverse Events by System Organ Class and Preferred Term
- (6) Intensity of Drug-Related Treatment-Emergent Adverse Events by System Organ Class, and Preferred Term
- (7) Treatment-Emergent Adverse Events Leading to Study Drug Discontinuation by System Organ Class and Preferred Term
- (8) Drug-Related Treatment-Emergent Adverse Events Leading to Study Drug Discontinuation by System Organ Class and Preferred Term
- (9) Serious Treatment-Emergent Adverse Events by System Organ Class and Preferred Term
- (10) Serious Drug-Related Treatment-Emergent Adverse Events by System Organ Class and Preferred Term
- (11) Treatment-Emergent Adverse Events by System Organ Class and Preferred Term **Over Time**
- (12) Most Frequent Treatment-Emergent Adverse Events by System Organ Class and Preferred Term
- (13) Treatment-Emergent Adverse Events Corresponding to Liver Function Test Abnormalities by System Organ Class and Preferred Term
- (14) Drug-Related Treatment-Emergent Adverse Events Corresponding to Liver



C-TMPL-DO-801 29 of 58 **Template Number:** Page: 1.0 **Version Number: Effective Date:** 02 Apr 2014 erins of Use

This version replaces: **TMPL-104** 

**Template Title:** Statistical Analysis Plan (Legacy Takeda)

Function Test Abnormalities by System Organ Class and Preferred Term

- (15) Significant Treatment-Emergent Adverse Events by System Organ Class and **Preferred Term**
- (16) Drug-Related Significant Treatment-Emergent Adverse Events by System Organ **Class and Preferred Term**
- (17) Most Frequent Non Serious Treatment-Emergent Adverse Events by System Organ **Class and Preferred Term**

The frequency distribution will be provided according to the rules below. Number of subjects

- Summary tables other than (5), (6) and (11) A subject with multiple occurrences of TEAE within a SOC will be counted only once in that SOC. A subject with multiple occurrences of TEAE within a PT will be counted only once in that PT. Percentages will be based on the number of subjects in the safety analysis set.
- Summary tables for (5) and (6) A subject with multiple occurrences of TEAE within a SOC or a PT will be counted only once for the TEAE with the maximum intensity. Percentages will be based on the number of subjects in the safety analysis set.
- Summary table for (11) A subject with a TEAE that occurs in more than one interval is counted in all the intervals that the TEAE occurs. For each time interval, a subject with multiple occurrences of TEAE within a SOC or a PT will be counted only once in that SOC or PT. When calculating percentages for each time interval, the number of subjects at risk (ie, subjects who either have an exposure or have an occurrence of TEAE, during or after the corresponding time interval) will be used as the denominator. The number of subjects whose onset of any one of the TEAEs is within the time interval will be used as the numerator.
- Summary table for (12) Most frequent TEAEs refer to PTs whose percentages are at least 2% in any one of the treatment groups.
- , roperty of Takeda. For Summary table for (17) Most frequent non-serious TEAEs refer to PTs that are not serious whose percentages are at least 5% in any one of the treatment groups. If there are no PTs whose percentages exceed 5%, the threshold is lowered to 2%. When calculating the percentages for "Subjects With Any TEAEs", the number of subjects with at least one of these most frequent non-serious TEAEs will be used as the numerator.



**Template Number:** C-TMPL-DO-801 30 of 58 Page: **Version Number:** 1.0 ible Leims of Use **Effective Date:** 02 Apr 2014

This version replaces: **TMPL-104** 

**Template Title:** Statistical Analysis Plan (Legacy Takeda)

#### 7.4.2 Pretreatment Events and Adverse Events in the Healing Phase

#### 7.4.2.1 Displays of Pretreatment Events

Analysis Set: All Subjects Who Signed the Informed Consent Form

Analysis Variables: PTE

Analytical Methods: The following summaries will be provided using frequency distribution.

PTEs will be coded using the MedDRA and will be summarized using SOC and PT. SOC will

be sorted alphabetically and PT will be sorted in decreasing frequency.

(1) Pretreatment Events by System Organ Class and Preferred Term

(2) Serious Pretreatment Events by System Organ Class and Preferred Term

The frequency distribution will be provided according to the rules below.

Number of subjects

A subject with multiple occurrences of PTE within a SOC will be counted only once in that SOC. A subject with multiple occurrences of PTE within a PT will be counted only once in

that PT.

# 7.4.2.2 Displays of Adverse Events in the Healing Phase

All Subjects Who Entered the Healing Phase Analysis Set:

Analysis Variables: AE in the Healing Phase

Analytical Methods: The following summaries will be provided using frequency distribution.

AEs will be coded using the MedDRA and will be summarized using SOC and PT. SOC will

be sorted alphabetically and PT will be sorted in decreasing frequency.

(1) Adverse Events in the Healing Phase by System Organ Class and Preferred Term

(2) Serious Adverse Events in the Healing Phase by System Organ Class and Preferred

The frequency distribution will be provided according to the rules below.

Number of subjects

Property of Lakeda. A subject with multiple occurrences of AE within a SOC will be counted only once in that SOC. A subject with multiple occurrences of AE within a PT will be counted only once in that



**Template Number:** C-TMPL-DO-801 31 of 58 Page: icable rems of Use **Version Number:** 1.0 **Effective Date:** 02 Apr 2014

This version replaces: **TMPL-104** 

**Template Title:** Statistical Analysis Plan (Legacy Takeda)

#### 7.4.3 Laboratory and Other Safety Data

## 7.4.3.1 Laboratory Test Results

### Hematology and Serum Chemistry

Analysis Set: Safety Analysis Set

Analysis Variables: Hematology

Red Blood Cells ( $\times 10^{12}/L$ ) White Blood Cells ( $\times 10^{9}/L$ ) Hemoglobin (g/L)

Platelets ( $\times 10^9/L$ ) Hematocrit (%)

White Blood Cell Fractions (Neutrophils (%), Eosinophils (%), Basophils (%),

Monocytes (%), Lymphocytes (%))

Serum Chemistry

ALT (U/L) ALP (U/L) AST (U/L)

Total Bilirubin (µmol/L) GGT (U/L) Direct Bilirubin (µmol/L)

CK (CPK) (U/L) LDH (U/L) Albumin (g/L) Creatinine (µmol/L) Total Protein (g/L) BUN (mmol/L)

Uric Acid (mmol/L) Total Cholesterol (mmol/L) Triglycerides (mmol/L)

Potassium (mmol/L) Sodium (mmol/L) Glucose (mmol/L)

Magnesium (mmol/L) Calcium (mmol/L) Inorganic Phosphorus (mmol/L)

Chloride (mmol/L) Serum Iron (µmol/L) Vitamin  $B_{12}$  (pmol/L)

ALT, AST, Total Bilirubin, and Direct Bilirubin: Visit:

> Baseline, Week 2, Week 4, Week 6, Week 8, Week 12, Week 24 Variables other than ALT, AST, Total Bilirubin, and Direct Bilirubin:

Baseline, Week 4, Week 12, Week 24

Analytical Methods: For each variable, summaries (1) and (2) will be provided by treatment group. Property of Takedai.

For applicable variables, summaries (3) and (4) will be provided by treatment group.

#### (1) Summary of Laboratory Test Results and Change from Baseline by Visit

Descriptive statistics for observed values and changes from baseline (each post-baseline visit - baseline) will be provided for each visit.

#### (2) Summary of Shifts of Laboratory Test Results

Shift tables showing the number of subjects in each category at baseline and each postbaseline visit will be provided. For each laboratory test, the laboratory values will be classified as "Low", "Normal" or "High" relative to the normal reference range provided by the central laboratory. The shift tables will be based on these classifications.

#### (3) Number and Percentage of Subjects with Markedly Abnormal Values of Laboratory **Parameters**

Overall frequency distributions of MAV during maintenance phase will be provided. If a




**TMPL-104** This version replaces:

**Template Title:** Statistical Analysis Plan (Legacy Takeda)

> laboratory parameter has both lower and upper MAV criteria, analysis will be performed for each. Further details are given in Appendix.

(4) Number and Percentage of Subjects with Elevated Liver Enzyme Laboratory

**Parameters** 

Overall frequency distributions of elevated hepatic parameters during maintenance phase will be provided. Further details are given in Appendix.

#### Urinalysis

Analysis Set: Safety Analysis Set

[Neg, Trace, 30 mg/dL, 100 mg/dL, 300 mg/dL, >=2000 mg/dL] Analysis Variables: Protein

> [Neg, 100 mg/dL, 250 mg/dL, 500 mg/dL, 1000 mg/dL, >=2000 mg/dL] Sugar

Visit: Baseline, Week 4, Week 12, Week 24

Analytical Methods: The following summaries will be provided for each treatment group.

(1) Summary of Shifts of Urine Laboratory Test Results

Shift tables showing the number of subjects in each category at baseline and each post-

ISE ONLY S baseline visit will be provided.

### Serum Gastrin, Pepsinogen I/II

Analysis Set: Safety Analysis Set

Analysis Variables: Serum Gastrin (pmol/L)

Pepsinogen I (µg/L) Pepsinogen II (µg/L) Pepsinogen I/II Ratio

Baseline, Week 4, Week 12, Week 24 Visit:

Analytical Methods: The following summaries will be provided for each treatment group.

Property of Takedai. For (1) Summary of Serum Gastrin and Pepsinogen I/II Results

For each visit, descriptive statistics for observed values and changes from baseline (each

post-baseline visit - baseline) will be provided.



**Template Number:** C-TMPL-DO-801 33 of 58 Page: applicable rems of Use **Version Number:** 1.0 **Effective Date:** 02 Apr 2014

This version replaces: **TMPL-104** 

**Template Title:** Statistical Analysis Plan (Legacy Takeda)

#### 7.4.4 Vital Signs, Physical Findings, and Other Observations Related to Safety

### Vital Signs

Analysis Set: Safety Analysis Set Analysis Variables: Body Temperature (C)

> Systolic Blood Pressure (mmHg) Diastolic Blood Pressure (mmHg)

Pulse (bpm)

Visit: Baseline, Week 4, Week 12, Week 24

Analytical Methods: For each variable, summaries (1) and (2) will be provided by treatment group.

(1) Summary of Vital Signs Parameters and Change from Baseline by Visit Descriptive statistics for observed values and changes from baseline (each post-baseline

visit – baseline) will be provided for each visit.

(2) Number and Percentage of Subjects with Markedly Abnormal Values of Vital Signs **Parameters** 

Overall frequency distributions of MAV during maintenance phase will be provided. If a vital sign parameter has both lower and upper MAV criteria, analysis will be performed for each. Further details are given in Appendix.

#### 12-lead ECG

Analysis Set: Safety Analysis Set Analysis Variables: Heart Rate (bpm)

> RR Interval (msec) PR Interval (msec) QT Interval (msec) QTcF Interval (msec) QRS Interval (msec)

Interpretation ["Within Normal Limits",

> "Abnormal, Not Clinically Significant", "Abnormal, Clinically Significant"]

Visit: Baseline, Week 12, Week 24

Analytical Methods: For each variable other than interpretation, summary (1) will be provided by treatment group.

For applicable variables, summary (2) will be provided by treatment group. For interpretation, summary (3) will be provided by treatment group.

(1) Summary of ECG Parameters and Change from Baseline by Visit

Descriptive statistics for observed values and changes from baseline (each post-baseline visit – baseline) will be provided for each visit.

(2) Number and Percentage of Subjects with Markedly Abnormal Values of ECG **Parameters** 

Overall frequency distributions of MAV during maintenance phase will be provided. If an



C-TMPL-DO-801 34 of 58 **Template Number:** Page: **Version Number:** 1.0 **Effective Date:** 02 Apr 2014

This version replaces:

**Template Title:** 

#### (3) Summary of Shifts of ECG Parameters

Summary of Shifts of ECG Parameters
Shift tables showing the number of subjects in each category at baseline and each postbaseline visit will be provided.

Analysis for China
ects in China

#### 7.4.5 **Subgroup Analysis for China**

Analysis Population: Subjects in China

Subjects in Countries other than China

Analytical Methods: (1) The same analyses as those in section 7.2 to 7.4.4 will be conducted for the subjects in

China.

(2) The same analyses as those in section 7.2 to 7.4.4 will be conducted for the subjects in countries other than China.

7.4.6 Subgroup Analysis for Taiwan

Analysis Population: Subjects in Taiwan

Analytical Methods: (1) The same analyses as those in section 72 to 7.4.4 will be conducted for the subjects in

#### Subgroup Analysis for Safety Analysis Set Excluding Accidentally 7.4.7 **Unblinded Subjects**

Analysis Population: Safety Analysis Set Excluding the Accidentally Unblinded Subjects

Safety Analysis Set Excluding the Accidentally Unblinded Subjects in China

Safety Analysis Set Excluding the Accidentally Unblinded Subjects in Countries other than

China

Safety Analysis Set Excluding the Accidentally Unblinded Subjects in Taiwan

Analytical Methods: The same analyses as those in sections 7.4.1.1 and 7.4.1.2 ((1), (4) to (17)) will be conducted in the safety analysis set that excludes subjects who were accidentally unblinded due to IWRS

system error.

The same analyses will be conducted for the subjects in China and countries other than China.

The same analyses will be conducted for the subjects in Taiwan.

# Significance Level and Confidence Coefficient

Significance level: 5% (two-sided test)

Confidence coefficient: 95% (two-sided)



scribed of Use applicable Terms of Use applicable Term **Template Number:** C-TMPL-DO-801  **Version Number:** 

This version replaces:

**Template Title:** 

#### 7.4.9 Changes in the Statistical Analysis Plan

The changes from the original SAP (Version: 1, Date: 20 November 2015) to the amended SAP were described below with a rationale for changes provided.

#### Page 1, TITLE PAGE

#### **Existing Text**

PPD

#### **Revised Text**

PPD

#### **Rationale for Amendment**

The responsible person has been changed.

#### Page 2, Section 1.0 APPROVAL SIGNATURES

**Existing Text** 

PPD

Revised Text

# Rationale for Amendment

The Responsible persons have been changed for Biostatistics and Clinical Science. The Responsible person has not been needed for Pharmacovigilance.

#### Page 7, Section 4.1 PRIMARY OBJECTIVES

#### **Existing Text**

To demonstrate the non-inferiority of TAK-438 to Lansoprazole in the reduction of relapse of erosive esophagitis in subjects in the Maintenance Phase (24 weeks) in whom endoscopic healing of erosive esophagitis has been



This version replaces: TMPL-104

Template Title: Statistical Analysis Plan (Legacy Takeda)

confirmed after treatment with TAK-438 or a PPI, as well as to determine the clinically recommended dose of TAK-438 for maintenance therapy in erosive esophagitis.

### **Revised Text**

- To demonstrate the non-inferiority of TAK-438 to Lansoprazole in the reduction of relapse of erosive esophagitis in subjects in the Maintenance Phase (24 weeks) in whom endoscopic healing of erosive esophagitis has been confirmed after treatment with TAK-438 or a PPI.
- To determine the clinically recommended dose of TAK-438 for maintenance therapy in erosive esophagitis in whom endoscopic healing of erosive esophagitis has been confirmed after treatment with TAK-438 or a PPI.

#### **Rationale for Amendment**

The description has been revised in the protocol.

# Page 7, Section 4.2 SECONDARY OBJECTIVES

# **Existing Text**

To evaluate the efficacy of TAK-438 during the 12-week treatment and the safety of TAK-438 versus Lansoprazole in subjects in the Maintenance Phase (24 weeks) in whom endoscopic healing of erosive esophagitis has been confirmed after treatment with TAK-438 or a PPI.

#### **Revised Text**

- To evaluate the efficacy of TAK-438 during the first 12-weeks of treatment in the Maintenance Phase in subjects with endoscopically confirmed healed erosive esophagitis receiving TAK-438 or a PPI.
- <u>To evaluate</u> the safety of TAK-438 versus Lansoprazole in subjects in the Maintenance Phase (24 weeks) in whom endoscopic healing of erosive esophagitis has been confirmed after treatment with TAK-438 or a PPI.

# **Rationale for Amendment**

The description has been revised in the protocol.

# Page 7~8, Section 4.4 STUDY DESIGN

#### **Existing Text**

This is a phase <u>III</u>, multicenter, double-blind, parallel-group <u>comparative</u> study <u>of TAK-438 (10 mg or 20 mg) in subjects in whom endoscopic healing of erosive esophagitis has been confirmed with TAK-438 or following proton <u>pump inhibitor (PPI) treatment</u>, to demonstrate the non-inferiority of TAK-438 to Lansoprazole <u>in their maintenance treatment (6 months or 24 weeks) as well as</u> to determine the clinically recommended dose <u>for TAK-438</u> for maintenance therapy in erosive esophagitis.</u>

All subjects who have been confirmed on endoscopy to have healing of erosive esophagitis will be randomized at a 1.1.1 ratio to oral TAK-438 10 mg, 20 mg or Lansoprazole 15 mg once daily given in the Maintenance Phase lasting 24 weeks.

If relapse of erosive esophagitis has been endoscopically confirmed in any subject, the subject will complete the study at that time point (to be construed as "complete cases in the Maintenance Phase", regardless of the time point where relapse of disease is confirmed).

This study will be conducted at a total of around  $\underline{60}$  sites across Asia with an estimated total of  $\underline{200}$  subjects randomized to each treatment group totaling 600 for the study.



Template Number: C-TMPL-DO-801 

This version replaces: TMPL-104

Template Title: Statistical Analysis Plan (Legacy Takeda)

The study will consist of a Screening Phase of up to 28 days <u>followed by a Treatment Phase of up to 24 weeks.</u>
There will be 5 subject visits scheduled: the start of the Screening Phase (Visit 1), the start of the Treatment Phase (Visit 2), after 4 weeks of treatment (Visit 3), after 12 weeks of treatment (Visit 4), after 24 weeks of treatment (Visit 5), and a Follow-up phase.

<u>Dosing will commence on Day 1 after randomization at Visit 2 (after completion of all required assessments scheduled on the day 1).</u>

#### **Revised Text**

This is a phase 3, multicenter, <u>randomized</u> double-blind, parallel-group study to demonstrate the non-inferiority of TAK-438 (10 mg or 20 mg) to Lansoprazole 15 mg in preventing the recurrence of erosive esophagitis in subjects with endoscopically confirmed healing of erosive esophagitis. This study also aims to determine the clinically recommended dose of TAK-438 for maintenance therapy of erosive esophagitis.

This study is comprised of 2 treatment periods: An open-label, single-arm period in which subjects receive Lansoprazole 30 mg for up to 8 weeks (Healing Phase), and a double-blind, parallel-group period in which subjects are randomized at a 1:1:1 ratio to TAK-438 10 mg, 20 mg or Lansoprazole 15 mg once daily for up to 24 weeks (Maintenance Phase). To enroll in the study subjects must have ongoing erosive esophagitis or have completed Study TAK-438 303. Subjects with ongoing erosive esophagitis are required to undergo the Healing Phase. Once erosive esophagitis healing is confirmed by endoscopy, these subjects may be randomized to 1 of 3 treatments in the Maintenance Phase. Subjects with endoscopic-confirmed healing of erosive esophagitis following the completion of Study TAK-438 303 will be randomized into the Maintenance Phase without carrying out the open-label Healing Phase. Subjects who previously entered the study (prior to Protocol Amendment 06) after confirmation of healed erosive esophagitis following treatment with a proton pump inhibitor (termed "de novo" subjects) are no longer eligible to enter the study; any ongoing subjects may continue being treated in the Maintenance Phase. A schematic of the study design is included in Figure 4.a.

If relapse of erosive esophagitis has been endoscopically confirmed in any subject, the subject will complete the study at that time point (to be construed as "complete cases in the Maintenance Phase"), regardless of the time point where relapse of disease is confirmed.

This study will be conducted at a total of around <u>70</u> sites across Asia with an estimated total of <u>231</u> subjects randomized to each treatment group <u>during the Maintenance Phase</u> (totaling <u>693 subjects entering the Maintenance Phase</u> for the study).

The study will consist of a Screening Phase of up to 28 days duration (Visit 1), a Healing Phase (for those subjects with ongoing erosive esophagitis only) of 4 or 8 weeks duration (Visits 2<sub>HP</sub> and 3<sub>HP</sub>), followed by a Maintenance Phase of up to 24 weeks (Visits 2-8), and a Follow-up Period of up to 14 days duration. With the exception of the Follow-up (which will be carried out by phone), all visits will occur at the clinic. The total duration of treatment is up to 6 months (24 weeks) in subjects entering from Study TAK-438 303, and up to 8 months (32 weeks) in subjects entering the study with ongoing erosive esophagitis.

Subjects with ongoing erosive esophagitis: Subjects who have ongoing erosive esophagitis will enter the Healing Phase and administration of Lansoprazole 30 mg once daily will commence following the completion of all required assessments at Visit 2<sub>HP</sub>. Subjects will then undergo a visit at Week -4 (Visit 3<sub>HP</sub>), where the subject may undergo endoscopy to confirm healing of erosive esophagitis. This is an optional procedure where the decision to perform endoscopy is based on the investigator's clinical judgment of a subject's symptoms of healing. Subjects who do not show endoscopic healing at Visit 3<sub>HP</sub> may continue in the Healing Phase and undergo endoscopy at Day 1 (Visit 2). Subjects with endoscopically confirmed healing of erosive esophagitis at Week -4 or at Day 1 will be eligible to enter the Maintenance Phase. Where the results from clinical laboratory tests confirming eligibility for the Maintenance Phase at Week -4 are not immediately available, subjects should continue to receive Lansoprazole 30 mg for up to 14 days. Subjects healed at Day 1 should be immediately randomized. Subjects who do not have




Subjects with healed erosive esophagitis: Subjects with healed erosive esophagitis will undergo a randomization visit (Visit 2), and dosing for the Maintenance Phase will commence following the completion of all required assessments on Day 1. Visits will then occur at 2 week intervals after the initiation of treatment of proton pump inhibitor outside Study TAV 400 no longer eligible. no longer eligible to enter the study; any ongoing subjects may continue to be treated in the Maintenance Phase.

All subjects receiving TAK-438 must undergo a total of 8 weeks of LFT monitoring visits with visits occurring every 2 weeks. For subjects entering the Maintenance Phase of the current study within 7 days of completing Study TAK-438 303, the requirement for 8 weeks of monitoring can be totalled across the 2 studies.

#### **Rationale for Amendment**

The descriptions have been revised in the protocol.

### Page 8, Section 4.4 STUDY DESIGN

#### **Existing Figure**





Template Number: C-TMPL-DO-801 

This version replaces: TMPL-104

Template Title: Statistical Analysis Plan (Legacy Takeda)

#### **Revised Figure**



### **Rationale for Amendment**

The figure (Figure 4.a) has been revised in the protocol.

# Page 9, Section 5.0 ANALYSIS ENDPOINTS

### **Existing Text**

The secondary efficacy endpoint for this study is the rate of recurrence\* of erosive esophagitis during the 12 weeks of treatment in the Maintenance Phase. Safety endpoints for this study include adverse events, clinical laboratory test results, ECG, vital signs, serum gastrin and pepsinogen I/II levels.

# **Revised Text**

The secondary efficacy endpoint for this study is the rate of recurrence\* of erosive esophagitis during the <u>first 12</u> weeks of treatment in the Maintenance Phase. Safety endpoints for this study include adverse events (AEs), clinical laboratory test results, ECG, vital signs, serum gastrin and pepsinogen I/II levels.

# **Rationale for Amendment**

The description has been revised in the protocol.

# Page 10, Section 6.0 DETERMINATION OF SAMPLE SIZE

### **Existing Text**

Assuming that the true Week 24 recurrence rate is 30.4% for <a href="lansoprazole">lansoprazole</a>, 22.0% for TAK-438 10 mg, and 13.6% for TAK-438 20 mg, and assuming that the dropout rate is <a href="up to 20%">up to 20%</a>, a sample size of <a href="185">185</a> subjects per group will provide an overall power of 90% to establish non-inferiority using a 2-sided 95% CI with a 10% non-inferiority margin. <a href="200">200</a> subjects per group will be included to allow adequate numbers for the regulatory requirements of various countries.



C-TMPL-DO-801 40 of 58 Template Number: Page: **Version Number:** 1.0 **Effective Date:** 02 Apr 2014

This version replaces: **TMPL-104** 

**Template Title:** Statistical Analysis Plan (Legacy Takeda)

The assumption of the true recurrence rate is based on a Phase 3 study that showed a Week 24 recurrence rate of 30.4% for lansoprazole 15 mg and 13.6% for lansoprazole 30 mg.

erms of Use Based on results from an earlier study of Lansoprazole as maintenance therapy for erosive esophagitis (AG-1749/CCT-202), the point estimate for the difference (Lansoprazole 15 mg group – Famotidine group) was calculated as -57.6% with the upper limit of the confidence interval being -30.7%. Therefore, the non-inferiority margin is specified as 10%.

### **Revised Text**

Assuming that the true Week 24 recurrence rate is 30.4% for Lansoprazole, 22.0% for TAK-438 10 mg, and 13.6% for TAK-438 20 mg, and assuming that the dropout rate is approximately 30%, a sample size of 208 subjects per group will provide an overall power of 90% to establish non-inferiority using a 2-sided 95% CI with a 10% noninferiority margin. 231 subjects per group will be included to allow adequate numbers for the regulatory requirements of various countries.

The assumption of the true recurrence rate is based on a phase 3 study that showed a Week 24 recurrence rate of 30.4% for Lansoprazole 15 mg and 13.6% for Lansoprazole 30 mg.

Based on results from an earlier study of Lansoprazole as maintenance therapy for erosive esophagitis (AG-1749/CCT-202), the point estimate for the difference (Lansoprazole 15 mg group – famotidine group) was calculated as -57.6% with the upper limit of the confidence interval being -30.7%. Therefore, the non-inferiority margin is specified as 10%.

#### Rationale for Amendment

The description with the targeted sample size has been revised in the protocol.


# **Existing Text**

TEAE: An adverse event whose date of onset occurs on or after the start of <u>study</u> drug.

# **Revised Text**

TEAE: An adverse event whose date of onset occurs on or after the start of the Maintenance Phase drug. A TEAE whose relationship to the Maintenance Phase drug is missing will be considered drug-related. A TEAE whose intensity is missing will be considered severe.

# **Rationale for Amendment**

The Maintenance Phase has been added in the protocol, and the handling rules for missing data for TEAE have been added.


### **Existing Text**

- Study Day: The day before the first dose of the study medication will be defined as Study Day -1 and the day of the first dose will be defined as Study Day 1. Other study days are defined relative to Study Day 1, eg, the day prior to Study Day 1 is Day -1 and the day after Study Day 1 is Day 2.
- Follow-up Day: The day after the last dose of the study medication will be defined as Follow-up Day 1. Other follow-up days are defined relative to Follow-up Day 1.



Template Number: C-TMPL-DO-801 

This version replaces: TMPL-104

Template Title: Statistical Analysis Plan (Legacy Takeda)

- Duration of exposure to study drug (days): date of last dose of study drug - date of first dose of study drug + 1

#### **Revised Text**

- Study Day: The day before the first dose of the <u>Maintenance Phase</u> drug will be defined as Study Day -1 and the day of the first dose will be defined as Study Day 1. Other study days are defined relative to Study Day 1, eg, the day prior to Study Day 1 is Day -1 and the day after Study Day 1 is Day 2.
- Follow-up Day: The day after the last dose of the <u>Maintenance Phase</u> drug will be defined as Follow-up Day 1. Other follow-up days are defined relative to Follow-up Day 1.
- Duration of exposure to study drug (days): date of last dose of <u>Maintenance Phase</u> drug date of first dose of <u>Maintenance Phase</u> drug + 1

#### **Rationale for Amendment**

The Maintenance Phase has been added in the protocol.


#### **Added Text**

Pepsinogen I/II Ratio: Pepsinogen I (µg/L) / Pepsinogen II (µg/L) (rounded to 1 decimal place)

Significant TEAE: Any TEAE (not including serious TEAEs) that led to an intervention, including withdrawal of drug treatment, dose increase, dose reduction or significant additional concomitant therapy.

#### **Rationale for Amendment**

The calculation formula for the above variable has been added with the number of decimal places. The significant TEAE should be analyzed and the definition of this type of TEAE has been added.

# Page 11~12, Section 7.1.2 Analysis Sets

# **Existing Text**

Analysis of efficacy variables will be conducted in the full analysis set (FAS) defined as all randomized subjects who receive at least 1 dose of <u>study medication</u> and have at least 1 post-baseline endoscopy, and will be based on the randomized treatment.

The primary efficacy endpoint and the secondary efficacy endpoint will also be analyzed in the per protocol set defined as all FAS subjects who did not have any of the major protocol deviations listed below. Analyses will be based on the randomized treatment.

- Subjects who did not meet inclusion criteria #3 or #4
- Subjects who met exclusion criteria #8, #11, #12, #13, or #14
- Subjects with study medication compliance of less than 70%
- Subjects who have been unblinded prior to database lock
- Subjects who have violated the rules specified in section 7.3 of the protocol

Analysis of safety variables will be conducted in the safety analysis set defined as all subjects who take at least 1 dose of <u>study medication</u> and will be based on the treatment received.



C-TMPL-DO-801 42 of 58 **Template Number:** Page: **Version Number:** 1.0 **Effective Date:** 02 Apr 2014

This version replaces: **TMPL-104** 

**Template Title:** Statistical Analysis Plan (Legacy Takeda)

#### **Revised Text**

Analysis of efficacy variables will be conducted in the full analysis set (FAS) defined as all randomized subjects who receive at least 1 dose of the Maintenance Phase drug and have at least 1 post-baseline endoscopy, and will be based on the randomized treatment. Randomized subjects who were accidentally unblinded due to IWRS system error will be excluded.

The primary efficacy endpoint and the secondary efficacy endpoint will also be analyzed in the per protocol set defined as all FAS subjects who did not have any of the major protocol deviations listed below. Analyses will be to the ap based on the randomized treatment.

- Subjects who did not meet inclusion criteria #3 or #4
- Subjects who met exclusion criteria #8, #11, #12, #13, or #14
- Subjects with study drug compliance of less than 70%
- Subjects who have been unblinded prior to database lock
- Subjects who have violated the rules specified in section 7.3 of the protocol

Analysis of safety variables will be conducted in the safety analysis set defined as all subjects who take at least 1 dose of the Maintenance Phase drug and will be based on the treatment received in the Maintenance Phase.

#### Rationale for Amendment

The Maintenance Phase has been added in the protocol. Accidental unblinding was identified in the study on Dec 16, 2015. It was confirmed that the treatment details of 93 subjects randomized in the study were accidentally unblinded to the site investigators, clinical project managers, and the CRA team through the IWRS subject visit notification emails. The accidental unblinding was caused by an WRS system error. The randomized subjects who were accidentally unblinded due to IWRS system error should be excluded from the FAS and the PPS.

# Page 12, Section 7.1.3 Handling of Rate of Endoscopic Recurrence of Erosive Esophagitis **Existing Text**

# 7.1.3.1 Rate of Endoscopic Recurrence of Erosive Esophagitis During the 12-Week Treatment

A subject who is diagnosed as LA classification grade A, B, C, or D from endoscopy tests performed between Study Day 2 and Study Day 127 (up to and including Follow-up Day 14) will be considered as a relapsed subject. Subjects who do not have any endoscopy data during this period will be treated as missing. Subjects who do not meet this requirement will be considered as 'not relapsed'. Recurrence rate will be calculated from the relapsed and not relapsed subjects, however, any subjects diagnosed as LA classification grade A, B, C, or D from endoscopy tests performed before the study medication administration will be excluded from the analysis.

# 7.1.3.2 Rate of Endoscopic Recurrence of Erosive Esophagitis During the 24-Week <u>Treatment</u>

A subject who is diagnosed as LA classification grade A, B, C, or D from endoscopy tests performed after Study Day 2 (up to and including Follow-up Day 14) will be considered as a relapsed subject. Subjects who do not have any endoscopy data during this period will be treated as missing. Subjects who do not meet this requirement will be considered as 'not relapsed'. Recurrence rate will be calculated from the relapsed and not relapsed subjects, however, any subjects diagnosed as LA classification grade A, B, C, or D from endoscopy tests performed before the study medication administration will be excluded from the analysis.



Template Number: C-TMPL-DO-801 

This version replaces: TMPL-104

Template Title: Statistical Analysis Plan (Legacy Takeda)

#### **Revised Text**

# 7.1.3.1 Rate of Endoscopic Recurrence of Erosive Esophagitis During the <u>first</u> 12 <u>Weeks of</u> Treatment <u>in the</u> Maintenance Phase

A subject who is diagnosed as LA classification grade A, B, C, or D from endoscopy tests performed between Study Day 2 and Study Day 127 (up to and including Follow-up Day 14) will be considered as a relapsed subject. Subjects who do not have any endoscopy data during this period will be treated as missing. Subjects who do not meet this requirement will be considered as 'not relapsed'. Recurrence rate will be calculated from the relapsed and not relapsed subjects, however, any subjects diagnosed as LA classification grade A, B, C, or D from endoscopy tests performed before the Maintenance Phase drug administration will be excluded from the analysis.

# 7.1.3.2 Rate of Endoscopic Recurrence of Erosive Esophagitis During the 24-Week Maintenance Phase

A subject who is diagnosed as LA classification grade A, B, C, or D from endoscopy tests performed after Study Day 2 (up to and including Follow-up Day 14) will be considered as a relapsed subject. Subjects who do not have any endoscopy data during this period will be treated as missing. Subjects who do not meet this requirement will be considered as 'not relapsed'. Recurrence rate will be calculated from the relapsed and not relapsed subjects, however, any subjects diagnosed as LA classification grade A, B, C, or D from endoscopy tests performed before the Maintenance Phase drug administration will be excluded from the analysis.

#### **Rationale for Amendment**

The Maintenance Phase has been added, and the description has been revised in the protocol.

# Page 12, Section 7.1.4 Handling of Data When Calculating Mean Severity According to Subject Diary

#### **Existing Text**

Mean severity = (total score of the severity recorded for the visit) / (number of days the severity of symptom is recorded) \*100 (rounded to 2 decimal places)

#### **Revised Text**

Mean severity = (total score of the severity recorded for the visit) / (number of days the severity of symptom is recorded) (rounded to 2 decimal places)

### Rationale for Amendment

The expression "\* 100" has been deleted because of clerical error.


#### **Existing Text**

Study Day: -28 - 1 (2 places)

#### Revised Text

Study Day: up to and including Study Day 1 (2 places)

# **Rationale for Amendment**

The time intervals should be changed because the Healing Phase has been added in the protocol.




# **Existing Text**

#### **Revised Text**

| ·<br>Version Number:<br>This version replaces:<br>Template Title: S | 1.0<br>TMPL-104<br>tatistical Analysis Plan (Legacy Tak | Effective Date | e: 02 Apr 201 | 4 |
|---|---|---|---|---|
| age 15, Section 7.1.6 Hand | lling of Other Endpoints | | | |
| xisting Text | | | | ins |
| linical laboratory tests, Gas | trin, Pepsinogen I/II, Vital signs | | ~ | |
| Version Number: 1.0 Effective Date: 02 Apr 2014 This version replaces: TMPL-104 Template Title: Statistical Analysis Plan (Legacy Takeda) age 15, Section 7.1.6 Handling of Other Endpoints xisting Text linical laboratory tests, Gastrin, Pepsinogen I/II, Vital signs evised Text linical laboratory tests (ALT, AST, total bilirubin, and direct bilirubin) | | | | |
| <u>Visit</u> | Scheduled Study Day | Time Int | erval (days) | |
| <u>v isit</u> | (days) | Study Day | Follow-up Day | |
| Baseline* | Study Day: 1 | <u>-28 – 1</u> | | |
| Week 2 | Study Day: 15 | 2-22 | up to and including<br>Follow-up Day 14 | |
| Week 4 | Study Day 29 | 23 – 36 | up to and including<br>Follow-up Day 14 | |
| Week 6 | Study Day: 43 | <u>37 – 50</u> | up to and including<br>Follow-up Day 14 | |
| Week 8 | Study Day: 57 | <u>51 - 71</u> | up to and including<br>Follow-up Day 14 | |
| <u>Week 12</u> | Study Day: 85 | <u>72 – 127</u> | up to and including<br>Follow-up Day 14 | |
| Week 24 | Study Day: 169 | <u>128 – 211</u> | up to and including<br>Follow-up Day 14 | |

<sup>\*:</sup> For the clinical laboratory tests of the subjects who participated in the TAK-438 303 study, if the last study visit coincides with the first visit in the 305 study or if the subject was randomized in the 305 study within 7 days after completing the last visit in the 303 study, then the data obtained at the last visit can be used as the baseline data for the 305 study.

Clinical laboratory tests (other than ALT, AST, total bilirubin, and direct bilirubin), Gastrin, Pepsinogen I/II, Vital signs

# **Rationale for Amendment**

Visit 3 (Week 2), Visit 5 (Week 6) and Visit 6 (Week 8) has been added in the protocol for evaluating liver function tests (ALT, AST, total bilirubin, and direct bilirubin).


For the clinical laboratory tests, gastrin and pepsinogen I/II, for the subjects who participated in the TAK-438 303 study

### **Revised Text**

For the clinical laboratory tests, gastrin, and pepsinogen I/II of the subjects who participated in the TAK-438 303 study



Template Number: C-TMPL-DO-801 

This version replaces: TMPL-104

Template Title: Statistical Analysis Plan (Legacy Takeda)

#### **Rationale for Amendment**

The expression has been revised.

# Page 16, Section 7.2.1.2 Screen Failures

# **Existing Text**

Race [American Indian or Alaska Native, Asian, Black or African American, Native Hawaiian or Other Pacific Islander, White]

#### **Revised Text**

Race [American Indian or Alaska Native, Asian, Black or African American, Native Hawaiian or Other Pacific Islander, White, Multiple]

#### **Rationale for Amendment**

There have been subjects whose race were "Multiple".

# Page 16, Section 7.2.1.3 Subject Eligibility

# **Existing Text**

Primary Reason for Subject Not Being Eligible [Pretreatment Event/Adverse Event, Major Protocol Deviation, Lost to Follow-Up, Voluntary Withdrawal, Study Termination, Did Not Meet Entrance Criteria, Other]

# **Revised Text**

Primary Reason for Subject Not Being Eligible Pretreatment Event/Adverse Event, Major Protocol Deviation, Lost to Follow-Up, Voluntary Withdrawal, Study Termination, Did Not Meet Entrance Criteria, <u>Healing Phase Failure</u>, Other]

# **Rationale for Amendment**

The category "Healing Phase Failure" has been added.

# Page 17, Section 7.2.1.5 Disposition of Subjects

#### Evicting Toyt

Study Drug (5 places)

### **Revised Text**

Maintenance Phase Drug (5 places)

### **Rationale for Amendment**

The Maintenance Phase has been added in the protocol.




This version replaces: TMPL-104

Template Title: Statistical Analysis Plan (Legacy Takeda)

### Page 17, Section 7.2.1.5 Disposition of Subjects

# **Existing Text**

# (1) Disposition of Subjects

Frequency distributions will be provided for each treatment group and overall. When calculating percentages for the reasons for not being treated, the total number of subjects not treated by the <u>study</u> drug will be used as the denominator. When calculating percentages for the reasons for discontinuation of <u>study</u> drug, the total number of subjects who prematurely discontinued the <u>study</u> drug will be used as the denominator.

#### **Revised Text**

# (1) Disposition of Subjects

Frequency distributions will be provided for each treatment group and overall. When calculating percentages for the reasons for not being treated, the total number of subjects not treated by the <u>maintenance phase</u> drug will be used as the denominator. When calculating percentages for the reasons for discontinuation of <u>maintenance phase</u> drug, the total number of subjects who prematurely discontinued the <u>maintenance phase</u> drug will be used as the denominator.

# (2) Flow Chart of Subject Distribution

Flow chart will be provided.

#### **Rationale for Amendment**

The Maintenance Phase has been added in the protocol. The analysis for providing a flow chart has been added in this SAP.

# Page 18, Section 7.2.2.1 Summary of Demographics and Other Baseline Characteristics

#### **Existing Text**

Analysis Set: Randomized Set

# **Revised Text**

Analysis Set: Randomized Set, Full Analysis Set

# **Rationale for Amendment**

The analysis for the full analysis set has been added.

# Page 18, Section 7.2.2.1 Summary of Demographics and Other Baseline Characteristics

# **Existing Text**?

Race [American Indian or Alaska Native, Asian, Black or African American, Native Hawaiian or Other Pacific Islander, White]

### **Revised Text**

Race [American Indian or Alaska Native, Asian, Black or African American, Native Hawaiian or Other Pacific Islander, White, Multiple]

# **Rationale for Amendment**

There have been subjects whose race were "Multiple".



Phase and subject to the applicable Terms of Use

Only and subject to the applicable Terms of Use

Only and subject to the applicable Terms of Use

Only and subject to the applicable Terms of Use

Only and subject to the applicable Terms of Use

Only and subject to the applicable Terms of Use

Only and subject to the applicable Terms of Use

Only and subject to the applicable Terms of Use Ter **Template Number:** C-TMPL-DO-801  **Version Number:** 1.0

This version replaces: **TMPL-104** 

**Template Title:** Statistical Analysis Plan (Legacy Takeda)

# Page 20, Section 7.2.3.1 Study Drug Exposure and Compliance

# **Existing Text**

Analysis Set: Safety Analysis Set

#### **Revised Text**

Analysis Set: Safety Analysis Set, Full Analysis Set

#### **Rationale for Amendment**

The analysis for the full analysis set has been added.

# Page 20, Section 7.2.3.1 Study Drug Exposure and Compliance

# **Existing Text**

(1) Study Drug Exposure and Compliance

#### **Revised Text**

(1) Study Drug Exposure and Compliance in Maintenance Phase

### **Rationale for Amendment**

The Maintenance Phase has been added in the protocol.

# Page 21, Section 7.3.1 Primary Efficacy Endpoint

# **Existing Text**

Rate of Endoscopic Recurrence of Erosive Esophagitis During the 24-week Treatment (3 places)

# **Revised Text**

Rate of Endoscopic Recurrence of Erosive Esophagitis During the 24-week Maintenance Phase (3 places)

# **Rationale for Amendment**

The Maintenance Phase has been added in the protocol.

# Page 21~22, Section 7.3.2 Secondary Efficacy Endpoint

# **Existing Text**

Rate of Endoscopic Recurrence of Erosive Esophagitis During the 12-week Treatment (4 places)

# **Revised Text**

Rate of Endoscopic Recurrence of Erosive Esophagitis During the First 12 Weeks of Treatment in the Maintenance Phase (4 places)

### **Rationale for Amendment**

The Maintenance Phase has been added in the protocol and the description has been revised in the protocol.



C-TMPL-DO-801 48 of 58 **Template Number:** Page: and it is a state of the second of the secon 1.0 **Version Number: Effective Date:** 02 Apr 2014

This version replaces: **TMPL-104** 

**Template Title:** Statistical Analysis Plan (Legacy Takeda)

### Page 24, Section 7.3.3.3 Barrett's Mucosa

### **Existing Text**

Present (3 cm or greater)

#### **Revised Text**

Present (3 cm or Greater)

#### Rationale for Amendment

The expression "greater" has been replaced with "Greater" because of clerical error.

# Page 24~26, Section 7.3.4 Statistical/Analytical Issues

# **Existing Text**

Rate of Endoscopic Recurrence of Erosive Esophagitis During the 24-week <u>Treatment</u> (7 places) Rate of Endoscopic Recurrence of Erosive Esophagitis During the 12-week Treatment (7 places)

#### **Revised Text**

Rate of Endoscopic Recurrence of Erosive Esophagitis During the 24-week Maintenance Phase (7 places) Rate of Endoscopic Recurrence of Erosive Esophagitis During the First 12 Weeks of Treatment in the Maintenance Phase (7 places)

#### **Rationale for Amendment**

The Maintenance Phase has been added in the protocol and the description has been revised in the protocol.

# Page 25, Section 7.3.4.2 Handling of Dropouts or Missing Data

# Added Text

Values below the lower limit of quantification will be treated as zero when calculating the descriptive statistics. Values above the upper limit of quantification will be treated as the upper limit values when calculating the descriptive statistics.

#### Rationale for Amendment

The handling rules of values below the lower or upper limit values for calculating the descriptive statistics have been added.

# Page 27, Section 7.4.1.1 Overview of Treatment-Emergent Adverse Events

# **Added Text**

5) Relationship to Study Drug of Treatment-Emergent Adverse Events Leading to Study Drug Discontinuation (number of events, number and percentage of subjects)

11) Significant Treatment-Emergent Adverse Events (number of events, number and percentage of subjects)

#### **Rationale for Amendment**

The analyses for these types of TEAEs have been added.



**Template Number:** C-TMPL-DO-801 49 of 58 Page: 1.0 Plicable Leurns of Use **Version Number: Effective Date:** 02 Apr 2014

This version replaces: **TMPL-104** 

**Template Title:** Statistical Analysis Plan (Legacy Takeda)

Page 28, Section 7.4.1.2 Displays of Treatment-Emergent Adverse Events

**Existing Text** 

System Organ Class

**Revised Text** 

SOC

**Rationale for Amendment** 

The expression "System Organ Class" has been replaced with "SOC" for expression consistency.

# Page 28~29, Section 7.4.1.2 Displays of Treatment-Emergent Adverse Events

#### **Added Text**

(8) Drug-Related Treatment-Emergent Adverse Events Leading to Study Drug Discontinuation by System Organ Class and Preferred Term

(10) Serious Drug-Related Treatment-Emergent Adverse Events by System Organ Class and Preferred Term

(15) Significant Treatment-Emergent Adverse Events by System Organ Class and Preferred Term

(16) Drug-Related Significant Treatment-Emergent Adverse Events by System Organ Class and Preferred Term

(17) Most Frequent Non Serious Treatment-Emergent Adverse Events by System Organ Class and Preferred Term

### Summary table for (17)

Most frequent non-serious TEAEs refer to PTs that are not serious whose percentages are at least 5% in any one of the treatment groups. If there are no PTs whose percentages exceed 5%, the threshold is lowered to 2%. When calculating the percentages for "Subjects With Any TEAEs", the number of subjects with at least one of these most frequent non-serious TEAEs will be used as the numerator.

### **Rationale for Amendment**

The analyses for these types of TEAEs has been added.

### Page 30, Section 7.4.2 Pretreatment Events and Adverse Events in the Healing Phase

#### **Existing Text**

7.4.2 Pretreatment Events

### Revised Text

7.4.2 Pretreatment Events and Adverse Events in the Healing Phase

(omitted)

7.4.2.2 Displays of Adverse Events in the Healing Phase

All Subjects Who Entered the Healing Phase Analysis Set:

Analysis Variables: AE in the Healing Phase



Template Number: C-TMPL-DO-801 

This version replaces: TMPL-104

Template Title: Statistical Analysis Plan (Legacy Takeda)

Analytical Methods: The following summaries will be provided using frequency distribution.

AEs will be coded using the MedDRA and will be summarized using SOC and PT. SOC will

be sorted alphabetically and PT will be sorted in decreasing frequency.

(1) Adverse Events in the Healing Phase by System Organ Class and Preferred Term

(2) Serious Adverse Events in the Healing Phase by System Organ Class and Preferred Term

The frequency distribution will be provided according to the rules below.

Number of subjects

A subject with multiple occurrences of AE within a SOC will be counted only once in that SOC. A subject with multiple occurrences of AE within a PT will be counted only once in that PT.

# **Rationale for Amendment**

The Healing Phase has been added in the protocol and the analyses for adverse events in the Healing Phase have been added in this SAP.

# Page 31~33, Section 7.4.3 Laboratory and Other Safety Data, Section 7.4.4 Vital Signs, Physical Findings, and Other Observations Related to Safety

# **Existing Text**

treatment phase (4 places)

### **Revised Text**

maintenance phase (4 places)

#### **Rationale for Amendment**

The Maintenance Phase has been added in the protocol.

# Page 31, Section 7.4.3.1 Laboratory Test Results

### **Existing Text**

Visit: Baseline, Week 4, Week 12, Week 24

# **Revised Text**

Visit: ALT, AST, Total Bilirubin, and Direct Bilirubin:

Baseline, Week 2, Week 4, Week 6, Week 8, Week 12, Week 24

Variables other than ALT, AST, Total Bilirubin, and Direct Bilirubin:

Baseline, Week 4, Week 12, Week 24

# Rationale for Amendment

Visit 3 (Week 2), Visit 5 (Week 6) and Visit 6 (Week 8) has been added in the protocol for evaluating liver function tests (ALT, AST, total bilirubin, and direct bilirubin).



**Template Number:** C-TMPL-DO-801  applicable Terms of Use **Version Number:** 1.0 **Effective Date:** 02 Apr 2014

This version replaces: **TMPL-104** 

**Template Title:** Statistical Analysis Plan (Legacy Takeda)

# Page 32, Section 7.4.3.1 Laboratory Test Results (Serum Gastrin, Pepsinogen I/II)

# **Existing Text**

Pepsinogen I (mcg/L), Pepsinogen II (mcg/L)

### **Revised Text**

Pepsinogen I (µg/L), Pepsinogen II (µg/L)

#### **Rationale for Amendment**

The expression "mcg" has been replaced with "ug" for using more suitable expression.

# Page 33, Section 7.4.4 Vital Signs, Physical Findings, and Other Observations Related to Safety (Vital Signs)

# **Existing Text**

Body Temperature (°C)

### **Revised Text**

Body Temperature (C)

# **Rationale for Amendment**

The expression "°C" has been replaced with "C" for using more suitable expression.

# Page 33, Section 7.4.4 Vital Signs, Physical Findings, and Other Observations Related to Safety (12-lead ECG)

# **Existing Text**

12-lead ECG interpretations (3 places)

# **Revised Text**

interpretations (3 places)

### **Rationale for Amendment**

The expression "12-lead ECG" has been deleted for expression consistency with TFLs.

# Page 34, Section 7.4.5 Subgroup Analysis for China

# **Existing Text**

Analysis Population: Subjects in China

Analytical Methods: The same analyses as those in section 7.2 to 7.4 will be conducted for the subjects in China.

# **Revised Text**

Analysis Population: Subjects in China

Subjects in Countries other than China

Analytical Methods: (1) The same analyses as those in section 7.2 to 7.4.4 will be conducted for the subjects in

China.



C-TMPL-DO-801 52 of 58 Template Number: Page: 1.0 **Version Number: Effective Date:** 02 Apr 2014

This version replaces: **TMPL-104** 

**Template Title:** Statistical Analysis Plan (Legacy Takeda)

3DIE Terms of Use (2) The same analyses as those in section 7.2 to 7.4.4 will be conducted for the subjects in countries other than China.

#### Rationale for Amendment

The analyses for the underlined part have been added.

# Page 34, Section 7.4.6 Subgroup Analysis for Taiwan, Section 7.4.7 Subgroup Analysis for Safety Analysis Set **Excluding Accidentally Unblinded Subjects**

#### Added Text

7.4.6 Subgroup Analysis for Taiwan

Analysis Population: Subjects in Taiwan

Analytical Methods: (1) The same analyses as those in section 7.2 to 7.4.4 will be conducted for the subjects in

Taiwan.

# 7.4.7 Subgroup Analysis for Safety Analysis Set Excluding Accidentally Unblinded Subjects

Analysis Population: Safety Analysis Set Excluding the Accidentally Unblinded Subjects

Safety Analysis Set Excluding the Accidentally Unblinded Subjects in China

Safety Analysis Set Excluding the Accidentally Unblinded Subjects in Countries other than

China

Safety Analysis Set Excluding the Accidentally Unblinded Subjects in Taiwan

Analytical Methods: The same analyses as those in sections 7.4.1.1 and 7.4.1.2 ((1), (4) to (17)) will be conducted

in the safety analysis set that excludes subjects who were accidentally unblinded due to IWRS

system error.

The same analyses will be conducted for the subjects in China and countries other than China.

The same analyses will be conducted for the subjects in Taiwan.

### **Rationale for Amendment**

The analyses for the underlined part have been added.

# Page 34, Section 7.4.6 Significance Level and Confidence Coefficient

# **Existing Text**

Significance level: 5% (two-sided test)

Confidence coefficient: 95% (two-sided)

No statistical testing will be performed if there are less than 5 subjects.

### **Revised Text**

Significance level: 5% (two-sided test)

Confidence coefficient: 95% (two-sided)



**Template Number:** C-TMPL-DO-801  ble reims of Use **Version Number:** 1.0 **Effective Date:** 02 Apr 2014

**TMPL-104** This version replaces:

Statistical Analysis Plan (Legacy Takeda) **Template Title:** 

#### **Rationale for Amendment**

The analysis plan has been changed that statistical testing will be performed even if there are less than 5 subjects.

# Page 54, Section 8.0 REFERENCES

#### **Added Text**

Luo N, et. al. (2017) "Estimating an EQ-5D-5L Value Set for China", Value in Health, Volume 20(4): 662-669.

#### Rationale for Amendment

The above reference has been added.

Page 56, Section 9.1.1 Hematology, Serum Chemistry, Urinalysis, Vital Signs, and 12-lead ECG (except Upper only and subject **MAV Criteria of QTcF Interval)** 

# **Existing Text**

Body Temperature ( ${}^{\circ}$ C)

### **Revised Text**

Body Temperature (C)

### **Rationale for Amendment**

a "C".

Property of Takeda. For non-commercial. The expression "°C" has been replaced with "C" for using more suitable expression.




**TMPL-104** This version replaces:

**Template Title:** 

## 8.0

DeLong ER, et. al. (1988) "Comparing the areas under two or more correlated receiver operating characteristic curves: a nonparametric approach", Biometrics, Volume 44(3): 837-45.

Divine G, et al. (2013) "A review of analysis and sample size calculation."

Anesth Analg, Volume 117(3): 699-710

- Lehmann EL, et. al. (1975) "Nonparametrics: statistical methods based on ranks", Springer.
- Mason SJ, et. al. (2002) "Areas beneath the relative operating characteristics (ROC) and relative operating levels (ROL) curves: Statistical significance and interpretation", Quarterly Journal of the Royal Meteorological Society (128): 2145-2166.
- a-N . China", Va.
  . China", Va.
  and Bull

  Property of Takeda: For non-commercial use only and such O'Brien RG, et. al. (2006) "Exploiting the link between the Wilcoxon-Mann-Whitney test and a simple odds statistic", Proceedings of the Thirty-First Annual SAS Users Group International Conference.
  - Luo N, et. al. (2017) "Estimating an EQ-5D-5L Value Set for China", Value in Health, Volume 20(4): 662-669.



Template Number: C-TMPL-DO-801 

This version replaces: TMPL-104

Template Title: Statistical Analysis Plan (Legacy Takeda)

# 9.0 APPENDIX

# 9.1 CRITERIA FOR MARKEDLY ABNORMAL VALUES

# 9.1.1 Hematology, Serum Chemistry, Urinalysis, Vital Signs, and 12-lead ECG (except Upper MAV Criteria of QTcF Interval)

For each parameter, all evaluable data (ie, non-missing data) obtained up to Follow-up Day 14 will be classified as a MAV or not. The criteria in the table below will be used.

For each parameter and subject, classifications will be made according to the conditions i) to iii) provided below. The lower and the upper criteria will be considered separately.

- i) A subject with at least one evaluable data after baseline that meets the MAV criteria will be classified as a subject with MAV.
- ii) A subject who does not meet condition i) and has at least one evaluable data after baseline that doesn't meet the MAV criteria will be considered as a subject without MAV.
- iii) A subject who does not meet conditions i) or ii) will be excluded from the analysis of MAV for that parameter.

Hematology

| Parameter | MAV Criteria | |
|-----------------------------------------|----------------|----------------|
| raiametei | Lower Criteria | Upper Criteria |
| Red Blood Cells ( $\times 10^{12}/L$ ) | <0.8×LLN | >1.2×ULN |
| White Blood Cells (×10 <sup>9</sup> /L) | <0.5×LLN | >1.5×ULN |
| Hemoglobin (g/L) | <0.8×LLN | >1.2×ULN |
| Hematocrit (%) | <0.8×LLN | >1.2×ULN |
| Platelets (×10 <sup>9</sup> /L) | <75 | >600 |
| Neutrophils (%) | <0.5×LLN | >1.5×ULN |
| Eosinophils (%) | - | >2×ULN |
| Basophils (%) | - | >3×ULN |
| Monocytes (%) | - | >2×ULN |
| Lymphocytes (%) | <0.5×LLN | >1.5×ULN |

Serum Chemistry

| Parameter | MAV Criteria | |
|---------------------------|----------------|----------------|
| Farameter | Lower Criteria | Upper Criteria |
| ALT (U/L) | - | >3×ULN |
| ALP (O/L) | - | >3×ULN |
| AST (U/L) | - | >3×ULN |
| GGT (U/L) | - | >3×ULN |
| Total Bilirubin (µmol/L) | - | >34.2 |
| Direct Bilirubin (μmol/L) | - | >2×ULN |
| CK (CPK) (U/L) | - | >5×ULN |
| Albumin (g/L) | <25 | - |
| Total Protein (g/L) | <0.8×LLN | >1.2×ULN |
| Creatinine (µmol/L) | - | >177 |
| BUN (mmol/L) | - | >10.7 |



Template Number: C-TMPL-DO-801 

This version replaces: TMPL-104

Template Title: Statistical Analysis Plan (Legacy Takeda)

| Parameter | MAV Criteria | |
|----------------------------------|----------------|----------------|
| Parameter | Lower Criteria | Upper Criteria |
| Uric Acid (mmol/L) | - | >0.773 |
| Total Cholesterol (mmol/L) | - | >7.72 |
| Triglycerides (mmol/L) | - | >2.5×ULN |
| Glucose (mmol/L) | <2.8 | >19.4 |
| Potassium (mmol/L) | <3.0 | >6.0 |
| Sodium (mmol/L) | <130 | €150 |
| Magnesium (mmol/L) | < 0.5 | >1.2 |
| Calcium (mmol/L) | <1.75 | >2.88 |
| Inorganic Phosphorus (mmol/L) | < 0.52 | >2.00 |
| Chloride (mmol/L) | <75 | >126 |
| Vitamin B <sub>12</sub> (pmol/L) | <92 | - |

Vital Signs

| Parameter | MAV Criteria | |
|---------------------------------|----------------|----------------|
| Faranicici | Lower Criteria | Upper Criteria |
| Body Temperature (C) | <35.6 | >37.7 |
| Systolic Blood Pressure (mmHg) | <85 | >180 |
| Diastolic Blood Pressure (mmHg) | <50 | >110 |
| Pulse (bpm) | <50 | >120 |

12-lead ECG

| Parameter | MAV Criteria | |
|----------------------|----------------|----------------|
| Parameter | Lower Criteria | Upper Criteria |
| Heart Rate (bpm) | <50 | >120 |
| QT Interval (msec) | <=50 | >=460 |
| QTcF Interval (msec) | <=50 | - |

# 9.1.2 12-lead ECG (Upper MAV Criteria of QTcF Interval)

All evaluable data (ie, non-missing data) obtained up to Follow-up Day 14 will be classified as a MAV or not. The criteria in the table below will be used. Note that the observed value and the change from baseline used for classification should be measurements taken on the same day.

For each subject, classifications will be made according to the conditions i) to iii) provided below.

- A subject with at least one evaluable data after baseline that meets the MAV criteria will be classified as a subject with MAV.
- A subject who does not meet condition i) and has at least one evaluable data after baseline that meets any of the following will be considered as a subject without MAV.
  - Observed value is less than 450 msec and not missing.
  - Change from baseline is less than 30 msec and not missing, and observed value is less than 500 msec and not missing.
- iii) A subject who does not meet conditions i) or ii) will be excluded from the analysis of MAV.



Template Number: C-TMPL-DO-801 

This version replaces: TMPL-104

Template Title: Statistical Analysis Plan (Legacy Takeda)

| Doromotor | MAV Criteria | |
|---|---|---|
| Parameter Lower Criteria | | Upper Criteria |
| QTcF Interval (msec) | - | If either of the following conditions is met: • observed value >=500 • change from baseline >= 30 and observed value >=450 |

# 9.2 CRITERIA FOR ELEVATED LIVER ENZYME

All evaluable data (ie, non-missing data) obtained up to Follow-up Day 14 will be used to determine whether each criteria for elevated liver enzyme in the table below is met or not. If there is more than one parameter that need to be considered for a criteria, parameter measurements taken on the same day will be used. For each criteria and subject, classifications will be made according to the conditions i) to iii) provided below.

- A subject who met criteria (a) at least once after baseline will be considered to have met the criteria for elevated liver enzyme.
- ii) If condition i) is not met but if criteria (b) is met at least once after baseline, then the subject will be considered to have not met the criteria for elevated liver enzyme.
- iii) If neither i) nor ii) is met, then the subject will be excluded from the analysis for the criteria for elevated liver enzyme.

| Label Criteria for Elevato | | ed Liver Enzyme |
|---|---|---|
| Label | (a) Elevated | (b) Not Elevated |
| ALT > 3xULN | ALT is greater than 3 times the ULN | ALT is non-missing and less than or equal to 3 times the ULN |
| ALT > 5xULN | ALT is greater than 5 times the ULN | ALT is non-missing and less than or equal to 5 times the ULN |
| ALT > 8xULN | ALT is greater than 8 times the ULN | ALT is non-missing and less than or equal to 8 times the ULN |
| ALT > 3xULN<br>with Tbili > 2xULN | ALT is greater than 3 times the ULN and the total bilirubin is greater than twice the ULN | Either ALT is non-missing and less than or equal to 3 times the ULN, or the total bilirubin is non-missing and less than or equal to twice the ULN |
| AST > 3xULN | AST is greater than 3 times the ULN | AST is non-missing and less than or equal to 3 times the ULN |
| AST > 5xULN | AST is greater than 5 times the ULN | AST is non-missing and less than or equal to 5 times the ULN |
| AST > 8xULN | AST is greater than 8 times the ULN | AST is non-missing and less than or equal to 8 times the ULN |
| AST > 3xULN<br>with Tbili > 2xULN | AST is greater than 3 times the ULN and the total bilirubin is greater than twice the ULN | Either AST is non-missing and less than or equal to 3 times the ULN, or the total bilirubin is non-missing and less than or equal to twice the ULN |
| ALT or AST > 3xULN | Either ALT or AST is greater than 3 times the ULN | Both ALT and AST are non-missing and less than or equal to 3 times the ULN |



Template Number: C-TMPL-DO-801 

This version replaces: TMPL-104

Template Title: Statistical Analysis Plan (Legacy Takeda)

| Label | Criteria for Elevated Liver Enzyme | |
|---|---|---|
| Label | (a) Elevated | (b) Not Elevated |
| ALT or AST > 5xULN | Either ALT or AST is greater than 5 times the ULN | Both ALT and AST are non-missing and less than or equal to 5 times the ULN |
| ALT or AST > 8xULN | Either ALT or AST is greater than 8 times the ULN | Both ALT and AST are non-missing and less than or equal to 8 times the ULN |
| ALT or AST > 3xULN with Tbili > 2xULN | Either ALT or AST is greater than 3 times the ULN and the total bilirubin is greater than twice the ULN | If any of the following conditions is met: - Both ALT and AST are non-missing and less than or equal to 3 times the ULN Total bilirubin is non-missing and less than or equal to twice the ULN. |
| ALT and AST > 3xULN | Both ALT and AST are greater than 3 times the ULN | Either ALT is non-missing and less than or equal to 3 times the ULN, or AST is non-missing and less than or equal to 3 times the ULN |
| ALT and AST > 5xULN | Both ALT and AST are greater than 5 times the ULN | Either ALT is non-missing and less than or equal to 5 times the ULN, or AST is non-missing and less than or equal to 5 times the ULN |
| ALT and AST > 8xULN | Both ALT and AST are greater than 8 times the ULN | Either ALT is non-missing and less than or equal to 8 times the ULN, or AST is non-missing and less than or equal to 8 times the ULN |
| ALT and AST > 3xULN with Tbili > 2xULN | Both ALT and AST are greater than 3 times the ULN and the total bilirubin is greater than twice the ULN | If any of the following conditions is met: - ALT is non-missing and less than or equal to 3 times the ULN - AST is non-missing and less than or equal to 3 times the ULN - Total bilirubin is non-missing and less than or equal to twice the ULN |
| ALP > 3xULN | ALP is greater than 3 times the ULN | ALP is non-missing and less than or equal to 3 times the ULN |
| ALP > 3xULN<br>with ALT > 3xULN | Both ALP and ALT are greater than 3 time the ULN | Either ALP is non-missing and less than or equal to 3 times the ULN, or ALT is non-missing and less than or equal to 3 times the ULN |
| ALP > 3xULN<br>with AST > 3xULN | Both ALP and AST are greater than 3 times the ULN | Either ALP is non-missing and less than or equal to 3 times the ULN, or AST is non-missing and less than or equal to 3 times the ULN |

# ELECTRONIC SIGNATURES

| | | EEECTROTTIC DIGITALI CRED | |
|---|---|---|---|
| | Signed by | Meaning of Signature | Server Date (dd-MMM-yyyy HH:mm 'UTC') |
| Pi | PD | Biostatistics Approval | (dd-MMM-yyyy HH;mm 'UTC')<br>10-Jan-2019 00:39 UTC |
| | | Biostatistics Approval | 10-Jan-201 <b>9 02</b> :19 UTC |
| | | Clinical Science Approval | 11 <b>-Jan-201</b> 9 07:14 UTC |
| | Forhoniconnic | Biostatistics Approval Clinical Science Approval Clinical Science Approval | |
| | of skegio. | | |
| Property | | | |